## Janssen Research & Development

## **Statistical Analysis Plan**

A Prospective, Multicenter, Open-Label, Single-Arm, Phase 2 Study to Investigate the Safety, Tolerability and Pharmacokinetics of Selexipag in Children with Pulmonary Arterial Hypertension (PAH)Protocol: AC-065A203

Protocol AC-065A203; Amendment 7; Phase 2

ACT-293987/JNJ-67896049 (selexipag)

Status: Approved

Date: 2 May 2022

**Prepared by:** Janssen Research & Development, a division of Janssen Pharmaceutical NV

**Document No.:** EDMS-597620, 1.0

Compliance: The study described in this report was performed according to the principles of Good Clinical Practice (GCP).

## **Confidentiality Statement**

The information provided herein contains Company trade secrets, commercial or financial information that the Company customarily holds close and treats as confidential. The information is being provided under the assurance that the recipient will maintain the confidentiality of the information under applicable statutes, regulations, rules, protective orders or otherwise.

## **TABLE OF CONTENTS**

| TABL | LE OF CONTENTS | 2 |
|---|---|---|
| VERS | SION HISTORY | 4 |
| 1. | INTRODUCTION | 5 |
| 1.1. | Study Objectives | |
| 1.2. | Study Objectives Study Design S | |
| 2. | ANALYSIS DETAILS | 7 |
| <del></del><br>2.1. | Analysis Sets | |
| 2.2. | Study Analysis Periods | |
| 2.3. | Study Output Deliverable | |
| 2.4. | Baseline Definition | |
| 3. | PARTICIPANT AND TREATMENT INFORMATION | 10 |
| 3.1. | Demographics and Baseline Disease Characteristics | 10 |
| 3.2. | Participant Recruitment, Disposition and Study Completion/Withdrawal Information | 10 |
| 3.3. | Previous and Concomitant Therapies and PAH-Specific Medications | 11 |
| 3.4. | Protocol Deviations | |
| 3.5. | Extent of Exposure and Compliance | |
| 3.6. | Individual maximum tolerated dose(iMTD) | |
| 3.7. | Other Participant Information | |
| | SAFETY ANALYSIS | 14 |
| 4.1. | Adverse Events | |
| 4.2. | Clinical Laboratory Tests | 16 |
| 4.3. | TSH, Thyroid antibodies and T3 and T4 | |
| 4.4. | Pregnancy Test | 19 |
| 4.5. | Electrocardiograms | |
| 4.6. | Vital Signs | 20 |
| 4.7. | Sexual maturation (Tanner Stage) | |
| 4.8. | Physical examination | 21 |
| | EXPLORATORY EFFICACY ANALYSIS | |
| 5.1. | The Exploratory Endpoints | |
| 5.2. | Analysis of the Exploratory Efficacy Variables | 22 |
| 5.2.1. | | |
| 5.2.2. | | |
| 5.2.3. | | |
| 5.2.4. | | |
| 5.2.5. | Disease Progression/Clinical Worsening | 23 |
| 6. | OTHER ENDPOINTS | 24 |
| 7. | STATISTICAL METHODS, CONVENTIONS FOR DISPLAYS AND DECIMAL PRECISION | 25 |
| 8. | SUPPORTING DOCUMENTATION | |
| 8.1. | Appendix 1 List of Abbreviations | 28 |
| 8.2. | Appendix 2 Definitions of Adverse Events of Special Interest | 29 |

## **LIST OF IN-TEXT TABLES AND FIGURES**

| Table 1: | SAP Version History Summary | 4 |
|----------|-----------------------------|---|
| Table 2: | Study Analysis Set Usage | 8 |
| | Study periods definition | |

## **VERSION HISTORY**

**Table 1:** SAP Version History Summary

| SAP Version | Approval Date | Change | Rationale |
|---|---|---|---|
| Original SAP | 10 June 2020 | Not Applicable | Initial release |
| Amendment 1 | 11 August 2020 | See rationale | 1) Add outputs for COVID-19 related AEs. |
| | | | 2) Add more analysis for concomitant PAH- |
| | | | specific medications |
| | | | 3) Update AESI definitions and provide more |
| | | | details on AESI definitions as an appendix |
| | | | of SAP to align with selexipag program |
| | | | level AESI definitions: ie. Remove |
| | | | thrombocytopenia from anaemia AESI |
| | | | definition, add PVOD AESI and medication |
| | | | error and pregnancy. |
| | | | 4) Add definitions for persistent and recurrent |
| | | | AESIs and average annualized event rates |
| Amendment 2 | 02 May 2022 | See rationale | 1) Update the SAP based on Protocol Version |
| | | | 8, Amendment 7 to add optional PK Interim |
| | | | Analysis 3. |
| | | | 2) Add Week 16 CSR deliverable, including all |
| | | | participants having Week 16 assessment. |
| | | | 3) Remove the persistent TEAE definition as |
| | | | the team agree that no separate output is |
| | | | need for it |

#### 1. INTRODUCTION

The purpose of this study is to confirm the selexipag doses in children from  $\ge 2$  to < 18 years of age with PAH that led to an exposure similar to that in adult participants. The selection of the selexipag starting dose was based on a PK extrapolation from adults to pediatric participants. In addition, the safety and tolerability of selexipag in children from  $\ge 2$  to < 18 years of age are assessed.

This statistical analysis plan (SAP) contains definitions of analysis sets, derived variables, and statistical methods for the analysis of safety and exploratory efficacy and other endpoints.

The analyses of pharmacokinetic (PK) data, as well as PK and PK/PD modeling are not included in this document but described in separate analysis plans.

## 1.1. Study Objectives

## Primary:

• The primary objective of the study is to confirm the selexipag starting dose(s), selected based on pharmacokinetic (PK) extrapolation from adults, which leads to similar exposures as adult doses in children from ≥2 to <18 years of age with pulmonary arterial hypertension (PAH) by investigating the PK of selexipag and its active metabolite ACT-333679 in this population.

## Secondary:

• To evaluate the safety and tolerability of selexipag in children from ≥2 to <18 years of age with PAH.

### *Exploratory*:

- To explore the relationship between drug exposure at the individual maximum tolerated dose (iMTD) and 6-minute walk distance (6MWD) at each time point of assessment.
- To explore the relationship between drug exposure and N-terminal pro b-type natriuretic peptide (NT pro-BNP) at each time point of assessment.
- To explore the relationship between drug exposure and Echocardiography (Echo) variables at each time point of assessment.
- To explore the time to disease progression/clinical worsening from first study drug dose up to EOT + 7 days.

#### Other:

- To assess palatability of selexipag formulation at each time point of assessment using a 5-point facial hedonic scale.
- To assess acceptability of selexipag formulation at each time point of assessment using a 3-point categorical scale.

## 1.2. Study Design

This is a prospective, multi-center, open-label, single-arm, Phase 2 study. Approximately 60 participants will be enrolled in 3 different age cohorts (based on age at baseline/enrollment/Visit 2) to obtain at least 45 participants with evaluable PK profiles:

• Cohort 1: ≥12 to <18 years of age (approximately 20 enrolled participants to obtain at least 15 participants with evaluable PK profiles)

- Cohort 2: ≥6 to <12 years of age (approximately 20 enrolled participants to obtain at least 15 participants with evaluable PK profiles)
- Cohort 3: ≥2 to <6 years of age (approximately 20 enrolled participants to obtain at least 15 participants with evaluable PK profiles).

The starting dose is based on the body weight category of the participants, using the data from the population PK model in the GRIPHON/AC-065A302 study targeting the exposure observed in adult PAH participants at a starting dose of 200  $\mu$ g, taken orally, twice a day. The continuous relationship between dose and body weight is used to define body weight categories and starting dose for each body weight category such that – on average – the exposure (AUC  $_{\tau,ss,\ combined}$ ) will be comparable to that of a 70 kg adult but not exceeding the exposure of a 50 kg adult.

## Dosing scheme (by body weight) is defined as follows:

- 100 µg starting dose for participants with a body weight from ≥9 to <25 kg
- 150 µg starting dose for participants with a body weight from  $\geq$ 25 to  $\leq$ 50 kg
- 200 μg starting dose for participants with a body weight ≥50 kg

Selexipag is to be dosed twice daily (bid) and during the up-titration period of 12 weeks, it is recommended that the doses are increased weekly in increments equal to the starting dose until the participants reach their individual maximum tolerated dose (iMTD), or until the maximum dose corresponding to 8-fold that of the starting dose (based on their baseline weight category) is achieved.

The starting dose selection will be confirmed or adjusted after completion of each age cohort by updating the population PK model (interim and final PK analysis).

Enrollment started with both Cohort 1 and Cohort 2 (participants  $\geq$ 12 to <18 years, and  $\geq$ 6 to <12 years of age, respectively). After completion of PK assessments in at least 15 participants in Cohort 1 at Week 12, the dose-exposure relationship was established using a population PK model (interim analysis 1). Enrollment of Cohort 3 (children  $\geq$ 2 to <6 years of age) was started once the appropriate doses were confirmed by modelling and simulation in a second interim analysis of PK data from the children older than 6 years (i.e., Cohorts 1 and 2) and the confirmation that there was no safety concern based on IDMC reviews.

The PK data pooled from all 3 age cohorts will be modelled to allow dosing recommendations for all children  $\ge 2$  years of age. A final PK analysis will be prepared based on the overall PK and safety data up to Week 16 evaluation. The selection of the dosing regimen for the Phase 3 study will be based on the safety, tolerability, and PK results evaluated in the interim or final PK analysis (as applicable).

Participants who discontinue the treatment any time before the profile PK sampling day will be replaced within the age cohort.

### **Study Periods**

The study consists of the following consecutive periods:

**Screening period:** Lasts up to 42 days; starts with the signature of the informed consent and ends with the administration of the first study treatment dose.

**Treatment period:** Starts from the first dose of study treatment at Baseline/enrollment visit and ends on the day of the last dose of selexipag (End of Treatment [EOT]). This includes:

### • Up-titration period:

From the first dose of study treatment until the participant reaches individual maximum tolerated dose (iMTD). This period is estimated to last up to 12 weeks.

## • Maintenance period:

**After Week 12:** the participants will continue study treatment at the same dose up to Week 16.

After Week 16: study treatment will continue as long as it remains beneficial for the participant up to maximum of 5 years after last (Cohort 3) participant first visit.

**EOT visit:** this visit should be conducted within 1 week of the last dose of study treatment.

**Safety Follow-up period:** Starts on the day after the last dose of study treatment and ends about 30 days thereafter with a phone call that indicates the End of Study (EOS).

#### 2. ANALYSIS DETAILS

## 2.1. Analysis Sets

- Screened Analysis Set: Screened analysis set includes all participants who are screened and have a participant identification number.
- Full Analysis Set: Full analysis set includes all enrolled participants who were eligible to receive the study drug.
- Safety Analysis Set: Safety analysis set includes all participants included in Full Analysis Set who receive at least one dose of the study drug. Since all enrolled participants received at least one dose of study drug, the Full Analysis Set and Safety Analysis Set are the same in this study. For simplicity, the Safety Analysis Set will be used for all safety and efficacy analyses.
- Pharmacokinetic Analysis Set (PKS): PK analysis set comprises all participants included in the Safety Analysis Set who complied with the protocol sufficiently and did not deviate from the protocol in a way that might affect the PK outcome of the study. Criteria for sufficient compliance include exposure to treatment, availability of PK measurements, and absence of major protocol deviations that have an impact on the PK. Further details are provided in the PK and modeling analysis plan.

For all analyses, except the time to disease progression event, only the scheduled visits data will be used in summary outputs; both the scheduled and unscheduled visits data will be included in the listings.

The analysis set usage is summarized as following:

Table 2: Study Analysis Set Usage

| | Screened | Full | Safety | PK | PK |
|---|---|---|---|---|---|
| | Analysis | Analysis | Analysis | Analysis | |
| | Set | Set | Set | Set | |
| Participant disposition | X | X | X | | |
| Participant information (medical | | | X | | |
| history, concomitant medication, | | | | | |
| contraceptives) | | | | | |
| Participant information | | | X | | |
| (demographics, baseline | | | | | |
| characteristics, baseline disease | | | | | |
| characteristics) | | | | | |
| Treatment exposure, treatment | | | X | | |
| discontinuation, drug accountability | | | | | |
| and compliance, protocol deviation | | | | | |
| Safety analyses | | | X | | |
| Other endpoints analyses | | | X | | |
| PK analyses | | | | X | X |
| Efficacy exploratory analyses | | | X | | |
| Sensitivity Analysis, for Efficacy | | | X | | |
| exploratory analyses | | | | | |
| All listings for | X | X | X | | |
| disposition/Recruitment | | | | | |
| All listings for Participant | X | X | X | | |
| information | | | | | |
| All other Listings | | | X | | |

## 2.2. Study Analysis Periods

For each dosed participant, the screening, treatment and follow-up phases of the study will be structured as following:

Table 3: Study periods definition

| Period | Period Start | Period End |
|---|---|---|
| Screening | Starts with the signature of the informed consent form (ICF), may be as early as Day -42 | Prior to the administration of the first study treatment dose |
| Treatment | | |
| Up-Titration | the first dose of study treatment | the participant reaches their iMTD (iMTD for each participant is determined at Week 12, or EOT + 3 days in case of premature treatment discontinuation before Week 12) |
| Maintenance after<br>Week 12 to 16<br>(continue treatment at<br>same dose) | Day of Up-Titration end plus 1. | Up to Week 16 or EOT + 3 days in case of premature treatment discontinuation before Week 16 |

| Period | Period Start | Period End |
|---|---|---|
| Maintenance after<br>Week 16 | Day of Week 16 visit plus 1 EOT (up to 5 years after last participal first visit) | |
| EOT visit | This visit should be conducted within 1 week of the last dose of study treatment. The participant will then enter the Safety follow-up period. | |
| Safety follow-up | Day after EOT | EOS - Day of Safety follow-up Phone call (about 30 days after last dose) |

In case a participant drops out during a treatment period, the participant will have a Follow-Up period after the last applicable treatment period only if a Follow-Up visit was performed.

Each of these analysis periods is associated with a treatment. Treatments for the Screening and Follow-Up periods are defined as 'None (screening/follow-up)', respectively.

## 2.3. Study Output Deliverable

This SAP will be used for Final Analysis CSR, Canada Health Authority Submission and Week 16 CSR. The data used by these deliverables are described as follows:

The Data Presentation Plan (DPS) will describe the details regarding which analyses and outputs are created for which purpose.

| Outputs Deliverables | Analysis Coverage/Data to include/Cut point |
|---|---|
| Analysis for Canada Health Authority Submission | Data cut-off: 04MAY2020 |
| | Data extract: 05MAY2020 |
| | Outputs for efficacy and safety |
| Week 16 CSR | All available participants' data in all age cohorts when all enrolled participants have finished all required Week 16 assessments or discontinued earlier from study permanently. Outputs for efficacy and safety |
| Final Analysis CSR | All datasets<br>Outputs for efficacy and safety |

#### 2.4. Baseline Definition

<u>Baseline</u>: Baseline will be defined as the last non-missing assessment available prior to the first dose administration. Any unscheduled measurement performed before administration of study drug should also be used for determination of baseline across all the domains, as some tests may be repeated for confirmation.

### 3. PARTICIPANT AND TREATMENT INFORMATION

## 3.1. Demographics and Baseline Disease Characteristics

For all Safety Analysis Set participants, descriptive summary statistics will be provided for the following by age cohort, body weight and in the overall population, and listings by age cohort, country, site.

- Demographic and baseline characteristics: Age (year with decimal for month) at enrollment, Sex, Childbearing Potential for female participants, Race, Ethnicity, Weight (kg), Height (cm), and BMI (kg/m²).
  - Childbearing Potential and sexual activity for female participants at Screening (or eventually at re-screening) will be summarized together with the above demographics.
- Baseline disease characteristics:

From the 'PAH Etiology' eCRF module:

- o Etiology of PAH, association of PAH with congenital heart disease (CHD),
- o Date of first observed/assumed PAH symptoms (only for listing),
- o Time from first observed/assumed symptoms (days) (date of first observed/assumed PAH symptoms date of screening + 1),
- o Date of PAH diagnosis (only for listing),
- O Time from PAH diagnosis (days) (date of PAH diagnosis date of screening + 1).

From the 'WHO Functional Class' eCRF module:

Baseline WHO Functional Class.

From the 'Panama Functional Class for Pediatrics' eCRF module:

o Baseline Panama FC.

From the 'Right Heart Catheterization' eCRF module:

- o Date of Diagnosis of right heart catheterization (RHC),
- o Mean pulmonary arterial pressure (mPAP[mmHg]),
- o Pulmonary arterial wedge pressure (PAWP[mmHg]) (or LAP or LVEDP),
- o Pulmonary vascular resistance index (PVRi[Wood units x m<sup>2</sup>]).
- Medical history (previous and ongoing clinically significant diseases) investigator original terms and preferred terms coded using the latest implemented MedDRA version dictionary will be listed.

# 3.2. Participant Recruitment, Disposition and Study Completion/Withdrawal Information

To describe participant disposition, the number of participants screened will be presented, and in addition, the following will be tabulated:

- Number (and % based on the Screened Analysis Set) of screening failures (all screened participants who were not enrolled)
  - Reasons for failure (from the "Enrollment" eCRF module)

- Number (and % based on the Screened Analysis Set) of enrolled participants (from the "Enrollment" eCRF module)
- Number (and % based on the Full Analysis Set) of dosed participants (with at least one record in the "Study Treatment Log" eCRF module)
- Number (and % based on the Safety Analysis Set) of participants who prematurely discontinued the study drug (from the "Premature Discontinuation of Study Treatment" and "Study Treatment Log eCRF modules)
  - o Reasons for treatment discontinuation
- Number (and % based on the Safety Analysis Set) of participants who completed the study as per protocol (with completed EOS follow-up telephone call)
- Date and time of informed consent with the protocol version will be listed together with enrollment data (including reasons for not enrolling the participants) for all participants in the Screened Analysis Set.
- Unmet inclusion criteria and met exclusion criteria will be also listed for participants in the Screened Analysis Set.
- A participant listing of recruitment by country and center will be provided based on the Screened Analysis Set. In addition, for the same analysis set the number of participants recruited in each country and center (within country) will be tabulated.
- Study completion/Study premature discontinuations along with relevant reasons will also be listed for all Safety Analysis Set participants ("Study Discontinuation" eCRF modules).

For an individual participant, per protocol study completion is reached when the EOS follow-up telephone call is completed.

Participants who prematurely discontinued study treatment for any reason before completion of the last study visit phase will not be considered to have completed the study.

Check the details for prematurely discontinuation of study treatment in Protocol 5.1.9.

#### 3.3. Previous and Concomitant Therapies and PAH-Specific Medications

All medications recorded in the 'Previous/Concomitant Medication' eCRF pages will be coded to preferred term using the latest version of the WHO Drug code and Anatomic Therapeutic Chemical class code dictionaries.

**Previous medications** are any medication/therapy with end date prior to the study drug start date.

Concomitant medications are defined as any medication/therapy with start date missing, or start date prior to, or on, or after the first study drug dose date but before last study drug dose, and with end date after the first study drug dose date, or end date missing.

In general, **concomitant medications** during study treatment include all medications taken whilst the participant is on study treatment, regardless of whether the start of intake is before the start of study drug. Concomitant medications include therefore concomitant medications at baseline and concomitant new medications.

Previous and concomitant medications (regardless of being PAH-specific or not) will be summarized by previous/concomitant medications class and preferred term and will be ordered according to decreasing frequency overall.

In addition, concomitant PAH-specific medications at baseline (i.e., used on the same day as the first dose of study drug but excluding the cases in which the medication ended on the day of first study drug dose), will be summarized. In this summary, PAH-specific medications will be presented by preferred term and PAH-specific medication subgroup name (as defined below). Also, the proportions of participants who received none, 1, 2, and 3 or more PAH-specific concomitant medications at baseline will be included.

The following preferred terms will define PAH-specific medications (except study treatment): "Ambrisentan", "Bosentan" (including "Bosentan Monohydrate"), "Sitaxentan", "Macitentan", "Sildenafil" (including "Sildenafil Citrate"), "Tadalafil", "Vardenafil", "Udenafil", "Riociguat", "Iloprost", "Epoprostenol", "Treprostinil", "Beraprost".

All other medications will be classified as non-PAH-specific medication.

PAH-specific medications at baseline summary will be provided by preferred term with the following subgroup treatment categories:

- Treatment with Endothelin Receptor Agonist (ERA) monotherapy identified by the following preferred terms ("Ambrisentan" OR "Bosentan" OR "Sitaxentan" OR "Macitentan") AND NOT ("Sildenafil" OR "Tadalafil" OR "Vardenafil" OR "Udenafil") AND NOT "Riociguat".
- Treatment with phosphodiesterase type 5 (PDE-5) inhibitor monotherapy identified by the following preferred terms ("Sildenafil" OR "Tadalafil" OR "Vardenafil" OR "Udenafil") AND NOT ("Ambrisentan" OR "Bosentan" OR "Sitaxentan" OR "Macitentan") AND NOT "Riociguat".
- Treatment with combination of both ERAs and PDE-5 inhibitors identified by the following preferred terms ("Ambrisentan" OR "Bosentan" OR "Sitaxentan" OR "Macitentan") AND ("Sildenafil" OR "Tadalafil" OR "Vardenafil" OR "Udenafil") AND NOT "Riociguat".
- Treatment with prostacyclin/analogs (irrespective of treatment with ERAs or PDE-5 inhibitors or "Riociguat") identified by the following preferred terms "Iloprost" OR "Epoprostenol" OR "Treprostinil" OR "Beraprost" (it is expected to be rare as prostacyclin/analogs are not allowed to be co-administered according to the study protocol).

• Treatment with soluble guanylate cyclase stimulator (irrespective of ERAs or PDE-5 inhibitors or prostacyclin/analogs) – identified by the preferred term "Riociguat".

All medications/therapies will be listed together. A different flag will indicate if the medication is previous or concomitant respectively. Additionally, forbidden and PAH-specific medications will be flagged.

All summaries will be provided by age cohort and body weight group.

All PAH-related non-pharmacological interventions recorded on the dedicated eCRF form will be listed.

If missing end date or the medications ended on or after first dose date of the study drug, the medication will be classified as concomitant medication. If both start date and end date are missing, then this medication will be considered as both previous and concomitant medications.

#### 3.4. Protocol Deviations

Major protocol deviations and COVID-19 related deviations will be reported in the database.

A listing of participants with major protocol deviations will be provided as well as a listing with any COVID-19 related deviations, including all available details about these deviations.

Between visits, compliance is expected to be between 80% and 120%. Compliance values outside of this range will be considered as protocol deviations (see details in Protocol 5.1.7.2.).

## 3.5. Extent of Exposure and Compliance

Exposure data are taken from the "Study Treatment Log" eCRF module.

All data recorded will be listed, together with treatment exposure duration (weeks) derived as defined below. The listing will also display the body weight at baseline, as this parameter triggers the starting dose.

Treatment duration (days) is defined as date of last intake of study drug minus date of first intake of study drug plus 1. It includes therefore any possible treatment interruption.

The treatment exposure duration (days) takes account of periods of drug interruption. To calculate the treatment exposure duration per participant, the number of days the participant took no study treatment is subtracted from the treatment duration defined above.

The treatment exposure duration (weeks) will be then calculated by dividing the treatment exposure duration (days) by 7.

Treatment duration or treatment exposure duration (weeks) will be summarized as categorical data. The duration categories will be cumulative for <=4 weeks, <=8 weeks, <=12 weeks, <=16 weeks, <=52 weeks.

Study treatment compliance is based on study treatment accountability. Study treatment compliance will be calculated by site personnel at visits as indicated in the assessment schedule using the below formula and entered in the eCRF:

Compliance = 100 x (number of tablets dispensed – number of tablets returned) / Total number of tablets that should have been taken during the period\*

\*The period is defined as the number of days of treatment from the date of dispensation / start of study treatment until the next accountability visit. The number of tablets that should have been taken should be calculated on a participant basis, based on the investigator's prescription.

Study treatment compliance, reason of non-compliance will be summarized at each timepoint. Details of study treatment dispensing and accountability will be listed for each participant.

#### 3.6. Individual maximum tolerated dose(iMTD)

The iMTD is defined as the last dose received before the Week 12 visit (for participants who prematurely discontinued study drug) or the dose received on the day of the Week 12 visit (for participants who completed the 12-week up-titration period).

For each iMTD, the number and percentage of participants who reached this dose will be summarized by age cohort and body weight group categories ( $\geq 9$  to <25 kg,  $\geq 25$  to <50 kg,  $\geq 50$  kg) at baseline.

The iMTD reached for each participant will be indicated in the study drug administration listing.

#### 3.7. Other Participant Information

Contraceptive methods used by female participants who are of childbearing potential and heterosexually active (or who become heterosexually active at any time after enrollment), collected on a dedicated eCRF module, will be listed.

#### 4. SAFETY ANALYSIS

Safety and tolerability will be assessed throughout the study, from signing of the Informed Consent Form (ICF) until the participant's last study-related activity. The study will include the following evaluations of safety and tolerability: adverse events, clinical laboratory tests (including TSH, thyroid antibodies, T3, T4, pregnancy tests, Plasma NT pro-BNP), ECG, vital signs, growth (weight, height and BMI), sexual maturation (Tanner Stage), childbearing potential and physical examinations.

Unless otherwise specified, all safety analyses will be carried out descriptively (using the Safety Analysis Set) in the overall population, by age cohort and body weight group.

#### 4.1. Adverse Events

#### **Adverse Events and Treatment-Emergent Adverse Events**

- Summaries of below adverse event categories will be summarized according to the study periods *Up-Titration*, *Maintenance after Week 12*, *Maintenance after Week 16* as defined in Table 2.
- All reported adverse events with onset following the start of study treatment, or preexisting conditions that have worsened since baseline, will be defined as treatmentemergent (TEAE) and will be included in the analysis. TEAEs will be recorded up to EOT + 3 days.
- AEs will be analyzed by period, and the start or worsened date-time of the AEs will be used to determine the period the AE falls in.
- For each TEAE, the percentage of participants who have experienced at least 1 occurrence of the given event will be summarized by system organ class, preferred term, and age cohort.
- TEAEs will be tabulated by severity and relationship and will be summarized by system organ class, preferred term, and age cohort.
- Serious AEs and AEs occurring up to EOT + 3 days that lead to death, hospitalization, treatment discontinuation, dose reduction/interruption will be tabulated and listed.
- AEs that occur during screening and that start prior to first dosing will be included in data listings only.
- All reported adverse event terms will be coded with the latest available MedDRA dictionary version.
- COVID-19 related AEs will be listed.

## **Adverse Events of Special Interest(AESI):**

Adverse events of special interest (AESI) for this study have been defined in Appendix 2.

For each AESI category, the percentage of participants who have experienced at least 1 occurrence of the given event will be summarized by system organ class, dictionary derived preferred term, and age cohort.

AESIs will be also tabulated by severity and will be presented by treatment periods, age cohort, body weight and overall. AESIs will also be summarized by relationship to the study drug.

Number of recurrent AESIs will be counted as the total number of occurrences of any TEAEs, i.e., multiple occurrences for the same preferred term for the same participant will be counted multiple times. Average annualized event rate will be calculated as follows:

- 1) Calculate total number of recurrent TEAEs.
- 2) Calculate participant-years of treatment duration (sum of individual participant timeyears in a treatment group)
- 3) Average annualized event rate = (total number of recurrent TEAE) / (subject-years of treatment duration)

The prostacyclin-associated Treatment-Emergent Adverse Events will be summarized by age cohort and body weight group during study period separately.

## **Deaths**

All AEs leading to death occurring up to 3 days after end of treatment, will be listed.

## **Hospitalization**

All hospitalization data from Hospitalization and Adverse Event CRF page will be listed.

## 4.2. Clinical Laboratory Tests

The following laboratory parameters are evaluated:

- Hematology:
  - Hemoglobin (g/L)
  - Hematocrit (L/L)
  - $\circ$  Erythrocyte count (10 $^{9}/L$ )
  - $\circ$  Leukocyte count with differential counts (10 $^9$ /L)
  - $\circ$  Platelet count (10<sup>9</sup>/L)
- Clinical chemistry:
  - o Alanine aminotransferase (U/L)
  - o Aspartate aminotransferase (U/L)
  - Alkaline phosphatase (U/L)
  - Total and direct bilirubin (μmol/L)
  - Creatinine (μmol/L)
  - Creatinine clearance (mL/min)
  - o Serum urea nitrogen (mmol/L)
  - Uric acid (µmol/L)
  - o Glucose (mmol/L)
  - o Cholesterol, triglycerides (mmol/L)
  - o Sodium, potassium, chloride, calcium (mmol/L)
  - o Albumin (g/L)
  - o NT-pro BNP (pmol/L)
  - o TSH (mU/L)
  - o Free T3 and free T4 (pmol/L)
  - o Thyroid antibodies (U/mL)

In addition, local laboratory parameters might be available under certain circumstances and recorded in the CRF.

All recorded assessments, whether from central or local laboratory (including unscheduled) will be assigned to the most appropriate visit time points according to the best fitting time-window for that assessment

If data from a local laboratory and from the central laboratory are available for the same date, the central laboratory value will be used; if more than one valid assessment are available on the same timepoint window in the same lab, the mean value will be considered.

A laboratory test abnormality is defined as any value outside the normal range as provided by the laboratory. The direction of the abnormality (below or above the normal range) is indicated using 'H' and 'L', if applicable.

A marked (alert) laboratory test abnormality is defined as any value that fulfills the applicable condition listed in the table below for LL / HH (or LLL / HHH, respectively):

| Safety parameter | Marked Abnormally<br>Low Values | | Marked Abnormally High Values | |
|---|---|---|---|---|
| | LL | LLL | НН | ннн |
| | Hematology | | | |
| Hemoglobin (g/L) | < 100 | < 80 | Increase (> 20 g/L)<br>above ULN or above<br>baseline if baseline is<br>above ULN | Increase (> 40 g/L) above ULN or above baseline if baseline is above ULN |
| Hematocrit (L/L) | < 0.28 F<br>< 0.32 M | < 0.20 | > 0.55 F<br>> 0.60 M | > 0.65 |
| Erythrocyte count (10 <sup>9</sup> /L) | NA | NA | NA | NA |
| Leukocyte count with differential counts (109/L) | < 3.0 | < 2.0 | > 20.0 | > 100.0 |
| Platelet count (10 <sup>9</sup> /L) | < 75 | < 50 | > 600 | > 999 |
| | | Clinic | al chemistry | |
| AST (U/L) | NA | NA | > 3 ' ULN | > 5 ' ULN |
| ALT (U/L) | NA | NA | > 3 ' ULN | > 5 ' ULN |
| Alkaline phosphatase (U/L) | NA | NA | > 2.5 ′ ULN | > 5 ' ULN |
| Total bilirubin<br>(μmol/L) | NA | NA | > 2 ' ULN | > 5 ' ULN |
| Direct bilirubin (μmol/L) | NA | NA | > 2 ' ULN | > 5 ' ULN |
| Creatinine (µmol/L) | NA | NA | > 1.5 'ULN or<br>> 1.5 ' baseline if<br>baseline is above ULN | > 3 ' ULN or<br>> 3 ' baseline if baseline<br>is above ULN |
| Serum urea nitrogen | NA | NA | > 2.5 x ULN | > 5 x ULN |
| Glucose (mmol/L) | < 3.0 | < 2.2 | > 8.9 | > 13.9 |
| Sodium (mmol/L) | NA | < 130 | > 150 | > 155 |
| Potassium (mmol/L) | < 3.2 | < 3.0 | NA | > 6.0 |
| Calcium (mmol/L) | < 2.0 | < 1.75 | > 2.9 | > 3.1 |

ALT = alanine aminotransferase; AST = aspartate aminotransferase; F = female; M = male; ULN = upper limit of normal range.

Treatment-emergent marked laboratory abnormalities are defined as all marked laboratory abnormalities with onset after the study treatment start and up to EOT+3 days, that were not present at baseline or worsened during the course of the study. They will be analyzed on the Safety Analysis Set overall, by age cohort and body weight group.

For each category (i.e., LL, LLL, HH, HHH), treatment-emergent marked laboratory abnormalities are summarized for each laboratory variable overall, by age cohort and body weight group, displaying counts and percentages of participants with at least one marked treatment-emergent abnormality. Percentages are calculated by dividing the number of participants with at least one marked abnormality for the parameter under consideration by the number of participants with any post-baseline measurement.

The number of participants with laboratory abnormalities/marked abnormalities (any value outside the normal ranges for the laboratory) will be also tabulated as shift tables against baseline.

Absolute values and changes from baseline will be determined for each parameter and participant at the different timepoints of assessment and summarized overall, by age cohort and body weight group for the Safety Analysis Set. For graphs or tables with mean values, to account for changing reference ranges across age and gender, certain central and local laboratory values (Y<sub>ori</sub>) and their reference ranges (LLN<sub>ori</sub>, ULN<sub>ori</sub>) will be normalized as Y<sub>norm</sub> using a standard range (LLN, ULN) as follows:

$$Y_{norm} = LLN + \frac{(Y_{ori} - LLN_{ori})}{(ULN_{ori} - LLN_{ori})} \times (ULN - LLN)$$

If the value is negative after normalization, zero will be assigned.

The laboratory tests that require normalization and their standard ranges to be used are:

- TSH: 0.34 5.60 (mIU/L)
- Free T3: 4.5 7.8 (pmol/L)
- Free T4: 10 24 (pmol/L)
- Hemoglobin: 116 164 (g/L)
- Hematocrit: 0.34 0.48 (L/L)
- Erythrocyte count: 4.1 5.6 (10<sup>12</sup>/L)
- Leukocyte count: 3.80 10.70 (10<sup>9</sup>/L)
- Neutrophil count:  $1.65 8.15 (10^9/L)$
- Lymphocyte count: 0.95 5.25 (10<sup>9</sup>/L)
- Monocyte count:  $0.40 0.90 (10^9/L)$
- Monocyte/leukocyte: 4.0 7.0 (%)
- Eosinophil count:  $0.00 0.20 (10^9/L)$
- Eosinophil/leukocyte: 0.0 4.1 (%)
- Platelet count:  $140 400 (10^9/L)$
- Creatinine: 40 83 (µmol/L)
- Alkaline phosphatase: 31-110 (U/L)

• Alanine aminotransferase: 6-34 (U/L)

• Aspartate aminotransferase: 10-40 (U/L)

• Uric Acid: 137-404 (μmol/L)

Albumin: 33 - 47 (g/L)
Triglyceride: 0.44 - 1.40 (mmol/L)

Iriglyceride: 0.44 - 1.40 (mmol/L)
 Cholesterol: 3.23 - 5.48 (mmol/L)

All individual laboratory data will be listed and a separate listing for participants with laboratory abnormalities will also be provided, as well as a separate listing of participants with treatment-emergent marked laboratory abnormalities.

## 4.3. TSH, Thyroid antibodies and T3 and T4

In addition, TSH (mU/L), thyroid antibodies (U/mL), free T3 (pmol/L) and free T4 values (pmol/L) will be presented separately.

## 4.4. Pregnancy Test

Serum pregnancy test will only be performed at screening. Afterwards urine pregnancy test will be performed. All results, as recorded in the eCRF, will be listed.

## 4.5. Electrocardiograms

ECG will be evaluated by a central ECG service. All ECG data from scheduled and unscheduled visits will be listed.

The quantitative ECG variables up to EOT + 3 days that will be summarized are heart rate (bpm), RR interval (msec), PR interval (msec), QRS interval (msec), QT interval (msec), QTcB (msec) and QTcF (msec), the corrected QT (QTc) using Bazett's and Fridericia's methods, respectively. Values at all scheduled visits and changes from baseline (last value assessed before first study dose intake) over time will be summarized by parameter, time point, age cohort and body weight, and will be presented in figures as well.

In addition, QTcB and QTcF will also be summarized by age cohort and the following categories:

- Value  $\leq 450$  (normal)
- Value > 450 480
- Value  $> 480 \le 500$
- Value > 500
- Increase from baseline < 30
- Increase from baseline  $> 30 \le 60$
- Increase from baseline > 60
- Value > 480 and increase from baseline  $> 30 \le 60$
- Value > 480 and increase from baseline > 60

For Week 1 and Week 12, where two additional ECG assessments are done at 2H and 4H post-dose, only pre-dose data will be included in the overall analysis. In addition, separate analyses will be done with only Week 1 and Week 12 ECGs data, where values and change from pre-dose to post-dose at each visit will be summarized by parameter, abnormality category for QTcB/F, time

point, and age cohort. Furthermore, summary of QTcF/B abnormalities by category over time and shift tables will be provided for both the overall analysis and Week 1 & 12-focused analysis.

The qualitative ECG abnormal findings at study baseline will be summarized by age cohort and are defined as following:

- Atrioventricular Conduction 1st Degree Av Block
- Chamber Hypertrophy or Enlargement Left Atrial Abnormality
- Chamber Hypertrophy or Enlargement Left Ventricular Hypertrophy
- Chamber Hypertrophy or Enlargement Right Atrial Abnormality
- Chamber Hypertrophy or Enlargement Right Ventricular Hypertrophy
- Interpretation Abnormal
- Interpretation Not Evaluable
- Intraventricular-Intraatrial Conduction Incomplete Right Bundle Branch Block
- Intraventricular-Intraatrial Conduction Intraventricular Conduction Delay, Nonspecific
- Intraventricular-Intraatrial Conduction Left Posterior Fascicular Block
- Intraventricular-Intraatrial Conduction Right Bundle Branch Block
- ST Segment. T wave, and U wave QTc Prolongation
- ST Segment. T wave, and U wave St Depression
- ST Segment. T wave, and U wave T Wave Inversion
- Sinus Node Rhythms and Arrhythmias Sinus Bradycardia
- Sinus Node Rhythms and Arrhythmias Sinus Tachycardia
- Supraventricular Arrhythmias Ectopic Atrial Rhythm

**Treatment-emergent qualitative ECG abnormalities**, defined as any ECG abnormal finding assessed up to EOT + 3 days and reported by the central ECG reader that was not present at study baseline (last assessment before first study drug intake), will also be summarized by age cohort. ECG abnormalities will be also presented in figures.

## 4.6. Vital Signs

The vital signs parameters up to EOT + 3 days that will be analyzed are heart rate and blood pressure (systolic and diastolic). Position and location will only be listed.

Values and change from baseline over time will be summarized by parameter and time point, age cohort and be presented in figures as well.

All individual vital signs data will be listed.

#### **Body Weight and Height**

Height (m) (measured at Screening and Week 16) and weight (kg) data will be used in calculating the BMI.

BMI (kg/m<sup>2</sup>) will be calculated at each of these time-points. Before Week 16, BMI is calculated by using height from screening, and at Week 16 will be calculated by using height collected at

Week 16. After Week 16, BMI will be calculated from the height and weight collected at each visit.

Values and changes from baseline over time for weight, height and BMI will be summarized by age cohort and body weight group.

All individual height, weight and BMI data will be listed, and the growth curves will be presented for height, weight, and BMI as well.

## 4.7. Sexual maturation (Tanner Stage)

Sexual maturation of pediatric participants in long-term studies is assessed by using Tanner Stage.

Tanner stage is assessed in female participants  $\geq 8$  years of age and in male participants  $\geq 9$  years of age. For participants who enter the study below these ages sexual maturity assessments will start once they reach the ages of 8 or 9 years. Tanner stage assessment is stopped once full sexual maturation is reached.

Tanner stage data will be listed and summarized along with changes from baseline (Screening) over time.

## Females of Childbearing Potential Status Change

Childbearing potential status assessed at screening will be listed with participant information, while changes in the status assessed for female participants at later timepoints will also be listed.

## 4.8. Physical examination

All data will be listed.

#### 5. EXPLORATORY EFFICACY ANALYSIS

All exploratory efficacy analyses will be carried out on the Safety Analysis Set, and be performed as follows:

- In the overall population.
- By age cohort.
- By body weight group

The main exploratory analysis will be based on observed data, with no imputation rules. Sensitivity analyses will be performed by imputing missing values as appropriate.

## 5.1. The Exploratory Endpoints

The exploratory endpoints are the following:

- Change from Baseline/Enrollment up to each time point of assessment in modified New York Heart Association / WHO FC.
- Change from baseline up to each time point of assessment in exercise capacity, as measured by the 6-minute walk distance (6MWD).

- Change from baseline in Panama FC up to each time point of assessment.
- Percent of baseline in plasma NT pro-BNP at each time point of assessment.
- Change from baseline up to each time point of assessment in Echo variables (imaging and Doppler evaluation):
  - o Right ventricular systolic pressure.
  - o Tricuspid annular plane systolic excursion.
  - Pulmonary artery acceleration time.
  - o Left ventricular eccentricity index.
  - o Right atrial area index (from apical 4 chamber view).
  - o Tricuspid annular diameter (from apical 4 chamber view).
- Time to first of the following disease progression events occurring between first study drug dose and EOT + 7 days:
  - o Death (all causes)
  - o Atrial septostomy or Potts' anastomosis, or registration on lung transplant list
  - Hospitalization due to worsening PAH<sup>§</sup>
  - Clinical worsening\* of PAH defined as: Need for, or initiation of new PAH-specific therapy<sup>#</sup> or i.v. diuretics or continuous oxygen use AND at least one of the following:
    - Worsening in WHO FC, or
    - New occurrence or worsening of syncope (in frequency or severity as per medical judgment), or
    - New occurrence or worsening of at least two PAH symptoms (i.e., shortness of breath/dyspnea, chest pain, cyanosis, dizziness/ near syncope, or fatigue), or
    - New occurrence or worsening of signs of right heart failure not responding to oral diuretics

§excluding hospitalizations that are elective, routine or clearly attributable to appearance/worsening of comorbidities (e.g., pneumonia).

<sup>#</sup>e.g., ERA, PDE-5 inhibitor, prostanoids, prostacyclin receptor (IP receptor) agonist, soluble guanylate cyclase stimulator.

## 5.2. Analysis of the Exploratory Efficacy Variables

#### 5.2.1. Modified NYHA/WHO FC and Panama FC

At each time point, change from Baseline of assessment in modified NYHA/WHO FC and Panama FC will be classified as worsened (> baseline value), unchanged (= baseline value) or improved (< baseline value) and be summarized by age cohort and body weight group.

All data will be listed too by age cohort, site ID, participant ID and body weight group.

 $CONFIDENTIAL-FOIA\ Exemptions\ \overline{Apply}\ in\ U.S.$ 

<sup>\*</sup>worsening from baseline.

#### 5.2.2. 6MWD

The change from baseline will be summarized at each time point of assessment up to the timepoint, using descriptive statistics for continuous variables. Two-sided 95% CIs of the mean and median will also be provided.

All exercise capacity data as measured by 6MWD test will be listed.

## 5.2.3. Plasma NT pro-BNP

The percent of baseline (defined as (NT pro-BNP value at the timepoint / NT pro-BNP at baseline [Day 1]) x 100) will be summarized at each time point of assessment and up to the timepoint with at least 10 participants in the age cohort, using descriptive statistics for continuous variables. The resulting mean and two-sided 95% CIs will be inversely transformed using the exponential function to provide the geometric mean and corresponding two-sided 95% CIs.

All data will be listed for each participant.

## 5.2.4. Echo/Doppler (assessed & transferred centrally)

The following Echo/Doppler variables, analyzed centrally, will be listed.

- Right ventricular systolic pressure (RVSP)
- Tricuspid annular plane systolic excursion (TAPSE)
- Pulmonary artery acceleration time)
- Left ventricular eccentricity index (LVEI)
- Right atrial area index (RAI)
- Tricuspid annular diameter

For each variable the change from baseline to each time point assessment will be summarized. Descriptive statistics for continuous variables will be displayed and the two-sided 95% CIs of the mean will also be provided.

## 5.2.5. Disease Progression/Clinical Worsening

Predefined signs and symptoms of PAH evaluated post baseline by the investigator to standardize the assessment of clinical worsening/disease progression and recorded in the eCRF will be listed.

In case of syncope or at least 2 new or worsening signs/symptoms the investigator must report disease progression in the eCRF and perform further exams to determine the cause.

Based on 'Disease progression event summary' the following time to event endpoint will be determined: time to disease progression/clinical worsening from first study drug dose up to EOT + 7 days.

All events (reasons) are considered:

• Death (all causes).

- Atrial septostomy or Potts' anastomosis, or registration on lung transplant list
- Hospitalization due to worsening PAH (excluding hospitalizations that are elective, routine or clearly attributable to appearance/worsening of comorbidities (e.g., pneumonia))
- Clinical worsening (from baseline) of PAH is defined as: need for, or the initiation of new PAH-specific therapy (e.g., ERA, PDE-5 inhibitor, prostanoids, prostacyclin receptor (IP receptor) agonist, soluble guanylate cyclase stimulator) or i.v. diuretics or continuous oxygen use AND at least one of the following:
  - o Worsening in WHO FC, or
  - New occurrence or worsening of syncope (in frequency or severity as per medical judgment), or
  - New occurrence or worsening of at least two PAH symptoms (i.e., shortness of breath/dyspnea, chest pain, cyanosis, dizziness/ near syncope, or fatigue), or
  - New occurrence or worsening of signs of right heart failure not responding to oral diuretic

Deaths (all causes) not reported in "disease progression event summary" by the investigators will also be included in this analysis.

Event time is defined as the time elapsed from the first study drug administration to the day of the first occurrence of the event.

If the date of onset of the event is incomplete it is set to the lower limit, unless the lower limit is before the study treatment start date in which case it is set to the study treatment start date.

The number (and percentage) of participants reporting each type of event will be tabulated by age cohort, weight group and overall, for first event and for all events.

Participants who did not experience an event will have their event time censored at EOT + 7 days. The number of participants at risk, the number of participants censored and the number of participants with event will be displayed together with Kaplan Meier estimates.

This time to event endpoint will be also graphically presented as Kaplan Meier estimates with 2-sided 95% CIs at relevant time points (where the number of participants at risk is at least 10% of the total number of participants in the analysis set).

The type and date of disease progression event, as well as time to event, will be listed for all participants; as for the event type of "clinical worsening", components of worsening will also be included in the listing, based on "clinical worsening of PAH".

#### 6. OTHER ENDPOINTS

#### Palatability and Acceptability of selexipag

Palatability and Acceptability of selexipag formulation will be assessed.

Answers for each question in the palatability questionnaire for Caregivers/Site Personnel, assessed via 5-point facial hedonic scale, will be summarized with counts and percentages by timepoint.

Acceptability of the selexipag formulation will be assessed through a 3-point categorical scale as to whether the child swallowed the medication at visits indicated in the assessment schedule: for all participants, parent(s) or LAR(s) or study site personnel will be asked following the drug intake whether the child swallowed the medication:

- a. fully,
- b. partially,
- c. not at all.

Answers for each question in acceptability questionnaire will be summarized with counts and percentages by timepoint.

Palatability and acceptability will also be listed.

# 7. STATISTICAL METHODS, CONVENTIONS FOR DISPLAYS AND DECIMAL PRECISION

Unless otherwise specified, all listings will be provided by center and participant number within each age cohort. They will be sorted then by assessment date as appropriate.

Descriptive summary statistics will be provided in the overall population, by age cohort and body weight group.

In summaries for categorical data all participants in the analysis set will be accounted for with tables displaying the number of participants with missing data. The number and percentage of participants in each category will be tabulated by visit as a shift table against baseline.

Summaries for continuous variables will include basic descriptive statistics: mean, median, first and third quartiles, standard deviation and range (minimum and maximum). Mean and median will be displayed as 1 decimal place more than the individual values. The standard deviations (SDs) will be displayed as 1 additional decimal place beyond that of the mean. If a count is 0, the percentage (0%) should not be displayed. The 0 count will be displayed, but the corresponding percentage should be omitted. If the corresponding denominator for the count is also 0, a hyphen (-) should be displayed rather than a 0 count or NA, and the corresponding percentage should be omitted.

- The participant percentages (%) presented in tables will be 1 decimal place unless the sample sizes for the percentages are small enough to warrant presenting as integers. The standard SAS rounding option will be used. For those percentages that rounds to 0.0, along with the count > 0, we will display < 0.1. For those percentages that would round to 100.0, where the count is less than the denominator, we will display > 99.9.
- All dates to be presented in Date9. format, along with time, wherever applicable.

#### Handling of Missing or Incomplete Date and Time Fields

Conventions for handling incomplete and missing dates are provided below. 'Lower limit' and 'upper limit' refer to the minimum or maximum, respectively, of a possible date. For example, if the day is missing, the lowest limit is the first day of the given month and the upper limit is the last day of the given month. If the day and month are missing, the lower limit refers to the 1st January of the given year and the upper limit to the 31st December of the given year.

| Type of Date | Date is incomplete | Date is missing |
|---|---|---|
| Date of PAH<br>diagnosis | Lower limit | No replacement |
| AE resolution date | The earlier of the Upper limit and the end of study date | No replacement, considered ongoing at end of study |
| AE onset date | If the end date of the AE is not before the start of study drug, and if the study drug start falls in the range of possible dates, it is the study drug start date. In all the other cases, it is the lower limit | The earlier of the end date of the AE and the start of study drug |
| Concomitant<br>medication start<br>date | Lower limit | No replacement, the medication is considered to have started before the study |
| Concomitant<br>medication end<br>date | The earlier of the Upper limit and the end of treatment date | No replacement, considered ongoing at end of treatment |
| Death date | Last of the Lower limit and recorded study assessment dates | Last of the recorded study assessment dates |

Anomalous information for a date will be handled using the following rules prior to using the imputations mentioned above:

If the day part of a date is non-numeric or has an invalid value, then day will be considered as missing. For example, if date = 44Nov2000 then, as it isn't possible to have a 44th day of the month, the day will be considered missing.

If the month part of a date does not match that of the possible months, then it will be considered missing, and so will the accompanying day. For example, if date = 21ND99 then both day and month will be considered as missing.

If the year part of a date is non-numeric or has an invalid value, then the whole date will be considered as missing.

## **General Conventions:**

- Study treatments start date is the first day of intake of study treatment. It is derived as the first 'Treatment start date' after sorting in chronological order all records. It coincides with Study Day 1.
- Study treatment end date (EOT) is the last day of intake of study treatment. It is derived as the last 'Treatment end date' after sorting in chronological order all records.
- Starting dose is the dose given on study treatment start date.

Study Day refers to the number of days elapsed since the day of study treatment start, plus 1 (i.e., Study Day 1 is the day of study treatment start). For dates prior to treatment start, it is the negative number of days elapsed between the date under consideration and the day of study treatment start. Therefore, the study day is always different from 0

#### 8. SUPPORTING DOCUMENTATION

## 8.1. Appendix 1 List of Abbreviations

6MWD 6-minute walk distance

AUC Area under the plasma concentration-time curve

 $AUC_{\tau,ss}$  Area under the plasma concentration-time curve over one dosing interval at steady-state

AUC<sub>t,ss,combined</sub> Combined exposure over one dosing interval at steady-state

 $C_{max}$  Maximum plasma concentration  $C_{max,ss}$  Maximum concentration at steady state

CHD Congenital heart disease
CSR Clinical Study Report
ECG Electrocardiogram
Echo Echocardiography

eCRF electronic Case Report Form

EOS End-of-Study
EOT End-of-Treatment
EU European Union
FAS Full analysis set
FC Functional class

GRIPHON Prostacyclin (PGI2G) receptor agonist in Pulmonary arterial Hypertension

i.v. Intravenous(ly)

ICF Informed Consent Form

IDMC Independent Data Monitoring Committee iMTD Individual maximum tolerated dose

LAP Left atrium pressure

LAR Legally authorized representative LVEDP Left ventricular end-diastolic pressure

MedDRA Medical Dictionary for Regulatory Activities

mPAP Mean pulmonary arterial pressure

NT pro-BNP N-terminal pro b-type natriuretic peptide

NYHA New York Heart Association
PAH Pulmonary arterial hypertension
PAWP Pulmonary arterial wedge pressure

PDE-5 Phosphodiesterase type-5 PK Pharmacokinetic(s)

PKS Pharmacokinetic Analysis Set

PT Preferred term

PVOD Pulmonary veno-occlusive disease PVR Pulmonary vascular resistance PVRi Pulmonary vascular resistance index

rhc Right heart catheterization
SAE serious adverse event
SAP Statistical Analysis Plan
SBP Systolic blood pressure
SD Standard deviation
SIV Site initiation visit
SOC System Organ Class

TEAE Treatment-emergent adverse event
TESAE Treatment-emergent serious adverse event

 $\begin{array}{ll} T_{max} & Time \ at \ which \ C_{max} \ is \ observed \\ TSH & Thyroid-stimulating \ hormone \\ WHO & World \ Health \ Organization \\ \end{array}$ 

## 8.2. Appendix 2 Definitions of Adverse Events of Special Interest

## **Definitions of Adverse Events of Special Interest**

## **TABLE OF CONTENTS** GASTROINTESTINAL DISTURBANCES DENOTING INTESTINAL INTUSSUSCEPTION (MANIFESTED AS ILEUS OR OBSTRUCTION)......47 HYPERTHYROIDISM .......47 HYPOTENSION .......50 LIGHT-DEPENDENT NON-MELANOMA SKIN MALIGNANCIES.......50 MAJOR ADVERSE CARDIOVASCULAR EVENTS......51 MEDICATION ERRORS.......58 OPHTHALMOLOGICAL EFFECTS ASSOCIATED WITH RETINAL VASCULAR SYSTEM ........ 61 1.10 PREGNANCY 67 1.11 PULMONARY VENOOCCLUSIVE DISEASE ASSOCIATED WITH PULMONARY

#### Overview

This appendix defines the <u>Adverse Events of Special Interest</u> (AESI) used in the tables and listings produced for study AC-065A203.

The MedDRA coding dictionary version used is 22.1 for Canada Submission and a later version will be used for final CSR.

## 1 Definition for each category of AESI

#### 1.1 Anaemia

Cases reporting events of anaemia are retrieved from the safety database for analysis if they contain an event Preferred Term (PT) within the 'Haematopoietic erythropenia' Standardised MedDRA Query (SMQ) (broad scope), or the 'Haematopoietic cytopenias affecting more than one type of blood cell' SMQ (broad scope, with the exception of 2 unspecific PTs: 'blood disorder', 'blood count abnormal'), or if they contain an event with any MedDRA PT containing the text 'anaemia', i.e., any of the following MedDRA PTs:

**ANAEMIA** 

ANAEMIA FOLATE DEFICIENCY

ANAEMIA HEINZ BODY

ANAEMIA MACROCYTIC

ANAEMIA MEGALOBLASTIC

ANAEMIA NEONATAL

ANAEMIA OF CHRONIC DISEASE

ANAEMIA OF MALIGNANT DISEASE

ANAEMIA OF PREGNANCY

ANAEMIA POSTOPERATIVE

ANAEMIA PROPHYLAXIS

ANAEMIA SPLENIC

ANAEMIA VITAMIN B12 DEFICIENCY

ANAEMIA VITAMIN B6 DEFICIENCY

APLASIA PURE RED CELL

APLASTIC ANAEMIA

ASPIRATION BONE MARROW ABNORMAL

**AUTOIMMUNE ANAEMIA** 

AUTOIMMUNE APLASTIC ANAEMIA

AUTOIMMUNE HAEMOLYTIC ANAEMIA

AUTOSOMAL RECESSIVE MEGALOBLASTIC ANAEMIA

**BICYTOPENIA** 

BIOPSY BONE MARROW ABNORMAL

BLOOD INCOMPATIBILITY HAEMOLYTIC ANAEMIA OF NEWBORN

**BLOOD LOSS ANAEMIA** 

BLOOD LOSS ANAEMIA NEONATAL

**BONE MARROW DISORDER** 

BONE MARROW FAILURE

BONE MARROW INFILTRATION

BONE MARROW MYELOGRAM ABNORMAL

**BONE MARROW NECROSIS** 

CARDIAC HAEMOLYTIC ANAEMIA

COLD TYPE HAEMOLYTIC ANAEMIA

CONGENITAL ANAEMIA

CONGENITAL APLASTIC ANAEMIA

CONGENITAL DYSERYTHROPOIETIC ANAEMIA

COOMBS NEGATIVE HAEMOLYTIC ANAEMIA

COOMBS POSITIVE HAEMOLYTIC ANAEMIA

**CYTOPENIA** 

**DEFICIENCY ANAEMIA** 

ERYTHROBLAST COUNT ABNORMAL

ERYTHROBLAST COUNT DECREASED

ERYTHROID MATURATION ARREST

**ERYTHROPENIA** 

ERYTHROPOIESIS ABNORMAL

ERYTHROPOIETIN DEFICIENCY ANAEMIA

FEBRILE BONE MARROW APLASIA

FOETAL ANAEMIA

FULL BLOOD COUNT DECREASED

GELATINOUS TRANSFORMATION OF THE BONE MARROW

HAEMATOCRIT ABNORMAL

HAEMATOCRIT DECREASED

**HAEMATOTOXICITY** 

HAEMOGLOBIN ABNORMAL

HAEMOGLOBIN DECREASED

HAEMOLYTIC ANAEMIA

HAEMOLYTIC ANAEMIA ENZYME SPECIFIC

HAEMOLYTIC ICTEROANAEMIA

HAND AND FOOT SYNDROME SECONDARY TO SICKLE CELL ANAEMIA

HEREDITARY HAEMOLYTIC ANAEMIA

HEREDITARY SIDEROBLASTIC ANAEMIA

HEXOKINASE DEFICIENCY ANAEMIA

HYPERCHROMIC ANAEMIA

HYPOCHROMIC ANAEMIA

HYPOPLASTIC ANAEMIA

IMMUNE-MEDIATED CYTOPENIA

IRON DEFICIENCY ANAEMIA

LEUKOERYTHROBLASTIC ANAEMIA

**MELANAEMIA** 

MICROANGIOPATHIC HAEMOLYTIC ANAEMIA

MICROCYTIC ANAEMIA

MYELODYSPLASTIC SYNDROME

MYELODYSPLASTIC SYNDROME TRANSFORMATION

**MYELOFIBROSIS** 

MYELOID METAPLASIA

**MYELOSUPPRESSION** 

NEPHROGENIC ANAEMIA

NORMOCHROMIC ANAEMIA

NORMOCHROMIC NORMOCYTIC ANAEMIA

NORMOCYTIC ANAEMIA

**PANCYTOPENIA** 

**PANMYELOPATHY** 

PERNICIOUS ANAEMIA

PLASMABLAST COUNT DECREASED

PRIMARY MYELOFIBROSIS

PROERYTHROBLAST COUNT ABNORMAL

PROERYTHROBLAST COUNT DECREASED

PROTEIN DEFICIENCY ANAEMIA

PYRUVATE KINASE DEFICIENCY ANAEMIA

RED BLOOD CELL COUNT ABNORMAL

RED BLOOD CELL COUNT DECREASED

REFRACTORY ANAEMIA WITH AN EXCESS OF BLASTS

REFRACTORY ANAEMIA WITH RINGED SIDEROBLASTS

RETICULOCYTE COUNT ABNORMAL

RETICULOCYTE COUNT DECREASED

RETICULOCYTE PERCENTAGE DECREASED

RETICULOCYTOPENIA

SCAN BONE MARROW ABNORMAL

SICKLE CELL ANAEMIA

SICKLE CELL ANAEMIA WITH CRISIS

SIDEROBLASTIC ANAEMIA

SPHEROCYTIC ANAEMIA

SPUR CELL ANAEMIA

WARM TYPE HAEMOLYTIC ANAEMIA

### 1.2 Bleeding events

Cases including events denoting haemorrhage or GI haemorrhage are retrieved from the safety database for analysis if they contain an event PT within either of the following MedDRA SMQs(narrow scope): 'Haemorrhage terms (excl. laboratory terms)', or 'Gastrointestinal haemorrhage', i.e., any of the following MedDRA PTs:

ABDOMINAL WALL HAEMATOMA

ABDOMINAL WALL HAEMORRHAGE

ABNORMAL UTERINE BLEEDING

ABNORMAL WITHDRAWAL BLEEDING

ACHENBACH SYNDROME

ACUTE HAEMORRHAGIC LEUKOENCEPHALITIS

ACUTE HAEMORRHAGIC ULCERATIVE COLITIS

ADMINISTRATION SITE BRUISE

| ADMINISTRATION SITE HAEMATOMA |
|----------------------------------------|
| ADMINISTRATION SITE HAEMORRHAGE |
| ADRENAL HAEMATOMA |
| ADRENAL HAEMORRHAGE |
| ANAL FISSURE HAEMORRHAGE |
| ANAL HAEMORRHAGE |
| ANAL ULCER HAEMORRHAGE |
| ANASTOMOTIC HAEMORRHAGE |
| ANASTOMOTIC ULCER HAEMORRHAGE |
| ANEURYSM RUPTURED |
| ANGINA BULLOSA HAEMORRHAGICA |
| ANORECTAL VARICES HAEMORRHAGE |
| ANTICOAGULANT-RELATED NEPHROPATHY |
| ANTIPLATELET REVERSAL THERAPY |
| AORTIC ANEURYSM RUPTURE |
| AORTIC DISSECTION RUPTURE |
| AORTIC INTRAMURAL HAEMATOMA |
| AORTIC PERFORATION |
| AORTIC RUPTURE |
| APONEUROSIS CONTUSION |
| APPLICATION SITE BRUISE |
| APPLICATION SITE HAEMATOMA |
| APPLICATION SITE HAEMORRHAGE |
| APPLICATION SITE PURPURA |
| ARTERIAL HAEMORRHAGE |
| ARTERIAL INTRAMURAL HAEMATOMA |
| ARTERIAL PERFORATION |
| ARTERIAL RUPTURE |
| ARTERIOVENOUS FISTULA SITE HAEMATOMA |
| ARTERIOVENOUS FISTULA SITE HAEMORRHAGE |
| ARTERIOVENOUS GRAFT SITE HAEMATOMA |
| ARTERIOVENOUS GRAFT SITE HAEMORRHAGE |
| ASTRINGENT THERAPY |
| ATRIAL RUPTURE |
| AURICULAR HAEMATOMA |
| BASAL GANGLIA HAEMATOMA |
| BASAL GANGLIA HAEMORRHAGE |
| BASILAR ARTERY PERFORATION |
| BLADDER TAMPONADE |
| BLEEDING VARICOSE VEIN |
| BLOOD BLISTER |

CONFIDENTIAL – FOIA Exemptions Apply in U.S.

35

| BLOOD LOSS ANAEMIA |
|--------------------------------------------------|
| BLOOD URINE |
| BLOOD URINE PRESENT |
| BLOODY DISCHARGE |
| BLOODY PERITONEAL EFFLUENT |
| BONE CONTUSION |
| BONE MARROW HAEMORRHAGE |
| BRAIN CONTUSION |
| BRAIN STEM HAEMATOMA |
| BRAIN STEM HAEMORRHAGE |
| BRAIN STEM MICROHAEMORRHAGE |
| BREAST HAEMATOMA |
| BREAST HAEMORRHAGE |
| BROAD LIGAMENT HAEMATOMA |
| BRONCHIAL HAEMORRHAGE |
| BRONCHIAL VARICES HAEMORRHAGE |
| BULLOUS HAEMORRHAGIC DERMATOSIS |
| BURSAL HAEMATOMA |
| CARDIAC CONTUSION |
| CAROTID ANEURYSM RUPTURE |
| CAROTID ARTERY PERFORATION |
| CATHETER SITE BRUISE |
| CATHETER SITE HAEMATOMA |
| CATHETER SITE HAEMORRHAGE |
| CENTRAL NERVOUS SYSTEM HAEMORRHAGE |
| CEPHALHAEMATOMA |
| CEREBELLAR HAEMATOMA |
| CEREBELLAR HAEMORRHAGE |
| CEREBELLAR MICROHAEMORRHAGE |
| CEREBRAL ANEURYSM PERFORATION |
| CEREBRAL ANEURYSM RUPTURED SYPHILITIC |
| CEREBRAL ARTERIOVENOUS MALFORMATION HAEMORRHAGIC |
| CEREBRAL ARTERY PERFORATION |
| CEREBRAL CYST HAEMORRHAGE |
| CEREBRAL HAEMATOMA |
| CEREBRAL HAEMORRHAGE |
| CEREBRAL HAEMORRHAGE FOETAL |
| CEREBRAL HAEMORRHAGE NEONATAL |
| CEREBRAL MICROHAEMORRHAGE |
| CERVIX HAEMATOMA UTERINE |
| CERVIX HAEMORRHAGE UTERINE |

CONFIDENTIAL – FOIA Exemptions Apply in U.S.

36
CHEST WALL HAEMATOMA CHOROIDAL HAEMATOMA CHOROIDAL HAEMORRHAGE CHRONIC GASTROINTESTINAL BLEEDING CHRONIC PIGMENTED PURPURA CILIARY BODY HAEMORRHAGE COITAL BLEEDING COLONIC HAEMATOMA CONJUNCTIVAL HAEMORRHAGE CONTUSION **CORNEAL BLEEDING CULLEN'S SIGN** CYSTITIS HAEMORRHAGIC DEEP DISSECTING HAEMATOMA DIARRHOEA HAEMORRHAGIC DISSEMINATED INTRAVASCULAR COAGULATION DIVERTICULITIS INTESTINAL HAEMORRHAGIC DIVERTICULUM INTESTINAL HAEMORRHAGIC **DUODENAL OPERATION** DUODENAL ULCER HAEMORRHAGE DUODENAL VASCULAR ECTASIA **DUODENITIS HAEMORRHAGIC** EAR HAEMORRHAGE **ECCHYMOSIS ENCEPHALITIS HAEMORRHAGIC** ENTEROCOLITIS HAEMORRHAGIC EPIDURAL HAEMORRHAGE **EPISTAXIS EXSANGUINATION** EXTRA-AXIAL HAEMORRHAGE EXTRADURAL HAEMATOMA EXTRADURAL HAEMATOMA EVACUATION EXTRAVASATION BLOOD **EYE CONTUSION** EYE HAEMATOMA EYE HAEMORRHAGE EYELID BLEEDING **EYELID CONTUSION** EYELID HAEMATOMA FEMORAL ARTERY PERFORATION FEMORAL VEIN PERFORATION

CONFIDENTIAL – FOIA Exemptions Apply in U.S.

FOETAL-MATERNAL HAEMORRHAGE FOTHERGILL SIGN POSITIVE GASTRIC ANTRAL VASCULAR ECTASIA GASTRIC HAEMANGIOMA GASTRIC HAEMORRHAGE GASTRIC OCCULT BLOOD POSITIVE GASTRIC ULCER HAEMORRHAGE GASTRIC ULCER HAEMORRHAGE, OBSTRUCTIVE GASTRIC VARICES HAEMORRHAGE GASTRITIS ALCOHOLIC HAEMORRHAGIC **GASTRITIS HAEMORRHAGIC** GASTRODUODENAL HAEMORRHAGE GASTROINTESTINAL ANASTOMOTIC LEAK GASTROINTESTINAL ANGIECTASIA GASTROINTESTINAL HAEMORRHAGE GASTROINTESTINAL POLYP HAEMORRHAGE GASTROINTESTINAL ULCER HAEMORRHAGE GASTROINTESTINAL VASCULAR MALFORMATION HAEMORRHAGIC **GENITAL CONTUSION** GENITAL HAEMORRHAGE GINGIVAL BLEEDING **GRAFT HAEMORRHAGE** GREY TURNER'S SIGN HAEMANGIOMA RUPTURE **HAEMARTHROSIS HAEMATEMESIS HAEMATOCHEZIA HAEMATOCOELE HAEMATOMA** HAEMATOMA EVACUATION HAEMATOMA INFECTION HAEMATOMA MUSCLE HAEMATOSALPINX **HAEMATOSPERMIA HAEMATOTYMPANUM** HAEMATURIA HAEMATURIA TRAUMATIC **HAEMOBILIA HAEMOPERITONEUM** HAEMOPHILIC ARTHROPATHY HAEMOPHILIC PSEUDOTUMOUR

Status: Approved, Date: 2 May 2022

| HAEMOPTYSIS |
|-------------------------------------------|
| HAEMORRHAGE |
| HAEMORRHAGE CORONARY ARTERY |
| HAEMORRHAGE FOETAL |
| HAEMORRHAGE IN PREGNANCY |
| HAEMORRHAGE INTRACRANIAL |
| HAEMORRHAGE NEONATAL |
| HAEMORRHAGE SUBCUTANEOUS |
| HAEMORRHAGE SUBEPIDERMAL |
| HAEMORRHAGE URINARY TRACT |
| HAEMORRHAGIC ADRENAL INFARCTION |
| HAEMORRHAGIC ARTERIOVENOUS MALFORMATION |
| HAEMORRHAGIC ASCITES |
| HAEMORRHAGIC BREAST CYST |
| HAEMORRHAGIC CEREBRAL INFARCTION |
| HAEMORRHAGIC CYST |
| HAEMORRHAGIC DIATHESIS |
| HAEMORRHAGIC DISEASE OF NEWBORN |
| HAEMORRHAGIC DISORDER |
| HAEMORRHAGIC EROSIVE GASTRITIS |
| HAEMORRHAGIC GASTROENTERITIS |
| HAEMORRHAGIC HEPATIC CYST |
| HAEMORRHAGIC INFARCTION |
| HAEMORRHAGIC NECROTIC PANCREATITIS |
| HAEMORRHAGIC OCCLUSIVE RETINAL VASCULITIS |
| HAEMORRHAGIC OVARIAN CYST |
| HAEMORRHAGIC STROKE |
| HAEMORRHAGIC THYROID CYST |
| HAEMORRHAGIC TRANSFORMATION STROKE |
| HAEMORRHAGIC TUMOUR NECROSIS |
| HAEMORRHAGIC URTICARIA |
| HAEMORRHAGIC VASCULITIS |
| HAEMORRHOIDAL HAEMORRHAGE |
| HAEMOSTASIS |
| HAEMOTHORAX |
| HEAVY MENSTRUAL BLEEDING |
| HENOCH-SCHONLEIN PURPURA |
| HEPATIC HAEMANGIOMA RUPTURE |
| HEPATIC HAEMATOMA |
| HEPATIC HAEMORRHAGE |
| HEREDITARY HAEMORRHAGIC TELANGIECTASIA |

| HYPERFIBRINOLYSIS |
|---------------------------------------|
| НҮРНАЕМА |
| ILIAC ARTERY PERFORATION |
| ILIAC ARTERY RUPTURE |
| ILIAC VEIN PERFORATION |
| IMMUNE THROMBOCYTOPENIA |
| IMPLANT SITE BRUISING |
| IMPLANT SITE HAEMATOMA |
| IMPLANT SITE HAEMORRHAGE |
| INCISION SITE HAEMATOMA |
| INCISION SITE HAEMORRHAGE |
| INCREASED TENDENCY TO BRUISE |
| INDUCED ABORTION HAEMORRHAGE |
| INFERIOR VENA CAVA PERFORATION |
| INFUSION SITE BRUISING |
| INFUSION SITE HAEMATOMA |
| INFUSION SITE HAEMORRHAGE |
| INJECTION SITE BRUISING |
| INJECTION SITE HAEMATOMA |
| INJECTION SITE HAEMORRHAGE |
| INSTILLATION SITE BRUISE |
| INSTILLATION SITE HAEMATOMA |
| INSTILLATION SITE HAEMORRHAGE |
| INTERMENSTRUAL BLEEDING |
| INTERNAL HAEMORRHAGE |
| INTESTINAL HAEMATOMA |
| INTESTINAL HAEMORRHAGE |
| INTESTINAL VARICES HAEMORRHAGE |
| INTRA-ABDOMINAL HAEMATOMA |
| INTRA-ABDOMINAL HAEMORRHAGE |
| INTRACEREBRAL HAEMATOMA EVACUATION |
| INTRACRANIAL HAEMATOMA |
| INTRACRANIAL TUMOUR HAEMORRHAGE |
| INTRAOCULAR HAEMATOMA |
| INTRAPARTUM HAEMORRHAGE |
| INTRATUMOURAL HAEMATOMA |
| INTRAVENTRICULAR HAEMORRHAGE |
| INTRAVENTRICULAR HAEMORRHAGE NEONATAL |
| IRIS HAEMORRHAGE |
| JOINT MICROHAEMORRHAGE |
| JUGULAR VEIN HAEMORRHAGE |

KIDNEY CONTUSION LACRIMAL HAEMORRHAGE LARGE INTESTINAL HAEMORRHAGE LARGE INTESTINAL ULCER HAEMORRHAGE LARYNGEAL HAEMATOMA LARYNGEAL HAEMORRHAGE LIP HAEMATOMA LIP HAEMORRHAGE LIVER CONTUSION LOWER GASTROINTESTINAL HAEMORRHAGE LOWER LIMB ARTERY PERFORATION LYMPH NODE HAEMORRHAGE MALLORY-WEISS SYNDROME MEDIASTINAL HAEMATOMA MEDIASTINAL HAEMORRHAGE MEDICAL DEVICE SITE BRUISE MEDICAL DEVICE SITE HAEMATOMA MEDICAL DEVICE SITE HAEMORRHAGE **MELAENA** MELAENA NEONATAL **MENINGORRHAGIA MENOMETRORRHAGIA** MESENTERIC HAEMATOMA MESENTERIC HAEMORRHAGE MOUTH HAEMORRHAGE MUCOCUTANEOUS HAEMORRHAGE MUCOSAL HAEMORRHAGE MUSCLE CONTUSION MUSCLE HAEMORRHAGE MYOCARDIAL HAEMORRHAGE MYOCARDIAL RUPTURE NAEVUS HAEMORRHAGE NAIL BED BLEEDING NASAL SEPTUM HAEMATOMA NEONATAL GASTROINTESTINAL HAEMORRHAGE NEPHRITIS HAEMORRHAGIC NIPPLE EXUDATE BLOODY OCCULT BLOOD POSITIVE OCULAR RETROBULBAR HAEMORRHAGE OESOPHAGEAL HAEMORRHAGE OESOPHAGEAL INTRAMURAL HAEMATOMA

CONFIDENTIAL – FOIA Exemptions Apply in U.S.

| OESOPHAGEAL ULCER HAEMORRHAGE |
|--------------------------------------|
| OESOPHAGEAL VARICES HAEMORRHAGE |
| OESOPHAGITIS HAEMORRHAGIC |
| OMENTAL HAEMORRHAGE |
| OPTIC DISC HAEMORRHAGE |
| OPTIC NERVE SHEATH HAEMORRHAGE |
| ORAL BLOOD BLISTER |
| ORAL CONTUSION |
| ORAL MUCOSA HAEMATOMA |
| ORAL PURPURA |
| ORBITAL HAEMATOMA |
| ORBITAL HAEMORRHAGE |
| OSTEORRHAGIA |
| OVARIAN HAEMATOMA |
| OVARIAN HAEMORRHAGE |
| PALPABLE PURPURA |
| PANCREATIC HAEMORRHAGE |
| PANCREATIC PSEUDOCYST HAEMORRHAGE |
| PANCREATITIS HAEMORRHAGIC |
| PAPILLARY MUSCLE HAEMORRHAGE |
| PARANASAL SINUS HAEMATOMA |
| PARANASAL SINUS HAEMORRHAGE |
| PARATHYROID HAEMORRHAGE |
| PAROTID GLAND HAEMORRHAGE |
| PELVIC HAEMATOMA |
| PELVIC HAEMATOMA OBSTETRIC |
| PELVIC HAEMORRHAGE |
| PENILE CONTUSION |
| PENILE HAEMATOMA |
| PENILE HAEMORRHAGE |
| PEPTIC ULCER HAEMORRHAGE |
| PERICARDIAL HAEMORRHAGE |
| PERINEAL HAEMATOMA |
| PERIORBITAL HAEMATOMA |
| PERIORBITAL HAEMORRHAGE |
| PERIOSTEAL HAEMATOMA |
| PERIPARTUM HAEMORRHAGE |
| PERIPHERAL ARTERY ANEURYSM RUPTURE |
| PERIPHERAL ARTERY HAEMATOMA |
| PERITONEAL HAEMATOMA |
| PERIVENTRICULAR HAEMORRHAGE NEONATAL |

**PETECHIAE** PHARYNGEAL CONTUSION PHARYNGEAL HAEMATOMA PHARYNGEAL HAEMORRHAGE PITUITARY APOPLEXY PITUITARY HAEMORRHAGE PLACENTA PRAEVIA HAEMORRHAGE POLYMENORRHAGIA POST ABORTION HAEMORRHAGE POST PROCEDURAL CONTUSION POST PROCEDURAL HAEMATOMA POST PROCEDURAL HAEMATURIA POST PROCEDURAL HAEMORRHAGE POST TRANSFUSION PURPURA POST-TRAUMATIC PUNCTATE INTRAEPIDERMAL HAEMORRHAGE POSTMENOPAUSAL HAEMORRHAGE POSTPARTUM HAEMORRHAGE PREMATURE SEPARATION OF PLACENTA PROCEDURAL HAEMORRHAGE PROCTITIS HAEMORRHAGIC PROSTATIC HAEMORRHAGE PULMONARY ALVEOLAR HAEMORRHAGE PULMONARY CONTUSION PULMONARY HAEMATOMA PULMONARY HAEMORRHAGE PULMONARY HAEMORRHAGE NEONATAL PUNCTURE SITE BRUISE PUNCTURE SITE HAEMATOMA PUNCTURE SITE HAEMORRHAGE PURPURA **PURPURA FULMINANS** PURPURA NEONATAL PURPURA NON-THROMBOCYTOPENIC **PURPURA SENILE** PUTAMEN HAEMORRHAGE RADIATION ASSOCIATED HAEMORRHAGE RECTAL HAEMORRHAGE RECTAL ULCER HAEMORRHAGE RENAL ARTERY PERFORATION RENAL CYST HAEMORRHAGE RENAL HAEMATOMA

CONFIDENTIAL – FOIA Exemptions Apply in U.S.

Status: Approved, Date: 2 May 2022

| RENAL HAEMORRHAGE |
|----------------------------------------|
| RESPIRATORY TRACT HAEMORRHAGE |
| RESPIRATORY TRACT HAEMORRHAGE NEONATAL |
| RETINAL ANEURYSM RUPTURE |
| RETINAL HAEMORRHAGE |
| RETINOPATHY HAEMORRHAGIC |
| RETROPERITONEAL HAEMATOMA |
| RETROPERITONEAL HAEMORRHAGE |
| RETROPLACENTAL HAEMATOMA |
| RUPTURED CEREBRAL ANEURYSM |
| SCLERAL HAEMATOMA |
| SCLERAL HAEMORRHAGE |
| SCROTAL HAEMATOCOELE |
| SCROTAL HAEMATOMA |
| SCROTAL HAEMORRHAGE |
| SHOCK HAEMORRHAGIC |
| SKIN HAEMORRHAGE |
| SKIN NEOPLASM BLEEDING |
| SKIN ULCER HAEMORRHAGE |
| SMALL INTESTINAL HAEMORRHAGE |
| SMALL INTESTINAL ULCER HAEMORRHAGE |
| SOFT TISSUE HAEMORRHAGE |
| SPERMATIC CORD HAEMORRHAGE |
| SPINAL CORD HAEMATOMA |
| SPINAL CORD HAEMORRHAGE |
| SPINAL EPIDURAL HAEMATOMA |
| SPINAL EPIDURAL HAEMORRHAGE |
| SPINAL SUBARACHNOID HAEMORRHAGE |
| SPINAL SUBDURAL HAEMATOMA |
| SPINAL SUBDURAL HAEMORRHAGE |
| SPLEEN CONTUSION |
| SPLENIC ARTERY PERFORATION |
| SPLENIC HAEMATOMA |
| SPLENIC HAEMORRHAGE |
| SPLENIC VARICES HAEMORRHAGE |
| SPLINTER HAEMORRHAGES |
| SPONTANEOUS HAEMATOMA |
| SPONTANEOUS HAEMORRHAGE |
| STOMA SITE HAEMORRHAGE |
| STOMATITIS HAEMORRHAGIC |
| SUBARACHNOID HAEMATOMA |

| SUBARACHNOID HAEMORRHAGE |
|-------------------------------------|
| SUBARACHNOID HAEMORRHAGE NEONATAL |
| SUBCAPSULAR HEPATIC HAEMATOMA |
| SUBCAPSULAR RENAL HAEMATOMA |
| SUBCAPSULAR SPLENIC HAEMATOMA |
| SUBCHORIONIC HAEMATOMA |
| SUBCHORIONIC HAEMORRHAGE |
| SUBCLAVIAN ARTERY PERFORATION |
| SUBCLAVIAN VEIN PERFORATION |
| SUBCUTANEOUS HAEMATOMA |
| SUBDURAL HAEMATOMA |
| SUBDURAL HAEMATOMA EVACUATION |
| SUBDURAL HAEMORRHAGE |
| SUBDURAL HAEMORRHAGE NEONATAL |
| SUBENDOCARDIAL HAEMORRHAGE |
| SUBGALEAL HAEMATOMA |
| SUBGALEAL HAEMORRHAGE |
| SUBRETINAL HAEMATOMA |
| SUPERIOR VENA CAVA PERFORATION |
| TESTICULAR HAEMORRHAGE |
| THALAMUS HAEMORRHAGE |
| THIRD STAGE POSTPARTUM HAEMORRHAGE |
| THORACIC HAEMORRHAGE |
| THROMBOCYTOPENIC PURPURA |
| THROMBOTIC THROMBOCYTOPENIC PURPURA |
| THYROID HAEMORRHAGE |
| TONGUE HAEMATOMA |
| TONGUE HAEMORRHAGE |
| TONSILLAR HAEMORRHAGE |
| TOOTH PULP HAEMORRHAGE |
| TOOTH SOCKET HAEMORRHAGE |
| TRACHEAL HAEMORRHAGE |
| TRAUMATIC HAEMATOMA |
| TRAUMATIC HAEMORRHAGE |
| TRAUMATIC HAEMOTHORAX |
| TRAUMATIC INTRACRANIAL HAEMATOMA |
| TRAUMATIC INTRACRANIAL HAEMORRHAGE |
| TUMOUR HAEMORRHAGE |
| ULCER HAEMORRHAGE |
| UMBILICAL CORD HAEMORRHAGE |
| UMBILICAL HAEMATOMA |

| UMBILICAL HAEMORRHAGE |
|------------------------------------|
| UPPER GASTROINTESTINAL HAEMORRHAGE |
| URETERIC HAEMORRHAGE |
| URETHRAL HAEMORRHAGE |
| URINARY BLADDER HAEMATOMA |
| URINARY BLADDER HAEMORRHAGE |
| URINARY OCCULT BLOOD |
| URINARY OCCULT BLOOD POSITIVE |
| UROGENITAL HAEMORRHAGE |
| UTERINE HAEMATOMA |
| UTERINE HAEMORRHAGE |
| VACCINATION SITE BRUISING |
| VACCINATION SITE HAEMATOMA |
| VACCINATION SITE HAEMORRHAGE |
| VAGINAL HAEMATOMA |
| VAGINAL HAEMORRHAGE |
| VARICOSE VEIN RUPTURED |
| VASCULAR ACCESS SITE BRUISING |
| VASCULAR ACCESS SITE HAEMATOMA |
| VASCULAR ACCESS SITE HAEMORRHAGE |
| VASCULAR ACCESS SITE RUPTURE |
| VASCULAR ANASTOMOTIC HAEMORRHAGE |
| VASCULAR GRAFT HAEMORRHAGE |
| VASCULAR PSEUDOANEURYSM RUPTURED |
| VASCULAR PURPURA |
| VASCULAR RUPTURE |
| VEIN RUPTURE |
| VENOUS HAEMORRHAGE |
| VENOUS PERFORATION |
| VENTRICLE RUPTURE |
| VERTEBRAL ARTERY PERFORATION |
| VESSEL PUNCTURE SITE BRUISE |
| VESSEL PUNCTURE SITE HAEMATOMA |
| VESSEL PUNCTURE SITE HAEMORRHAGE |
| VITREOUS HAEMATOMA |
| VITREOUS HAEMORRHAGE |
| VULVAL HAEMATOMA |
| VULVAL HAEMATOMA EVACUATION |
| VULVAL HAEMORRHAGE |
| WHITE NIPPLE SIGN |
| WITHDRAWAL BLEED |

WOUND HAEMATOMA
WOUND HAEMORRHAGE

# 1.3 Gastrointestinal disturbances denoting intestinal intussusception (manifested as ileus or obstruction)

Cases including events denoting GI disturbances are retrieved from the safety database for analysis if they contain an event with any MedDRA PT containing the text 'ileus', 'intestinal obstruction', 'intestinal pseudo-obstruction', 'intussusception', or 'volvulus', with the exception of unspecific PT: 'keratomileusis', i.e., any of the following MedDRA PTs:

| CONGENITAL INTESTINAL OBSTRUCTION |
|--------------------------------------------|
| DISTAL INTESTINAL OBSTRUCTION SYNDROME |
| GALLBLADDER VOLVULUS |
| GALLSTONE ILEUS |
| GASTRIC ILEUS |
| GASTRIC VOLVULUS |
| GASTROINTESTINAL OBSTRUCTION |
| ILEUS |
| ILEUS PARALYTIC |
| ILEUS SPASTIC |
| INTESTINAL OBSTRUCTION |
| INTESTINAL PSEUDO-OBSTRUCTION |
| INTUSSUSCEPTION |
| LARGE INTESTINAL OBSTRUCTION |
| LARGE INTESTINAL OBSTRUCTION REDUCTION |
| MALIGNANT GASTROINTESTINAL OBSTRUCTION |
| MECHANICAL ILEUS |
| MECONIUM ILEUS |
| NEONATAL INTESTINAL OBSTRUCTION |
| POSTOPERATIVE ILEUS |
| SMALL INTESTINAL INTUSSUSCEPTION REDUCTION |
| SMALL INTESTINAL OBSTRUCTION |
| SMALL INTESTINAL OBSTRUCTION REDUCTION |
| SUBILEUS |
| VOLVULUS |
| VOLVULUS OF SMALL BOWEL |
| VOLVULUS REPAIR |

# 1.4 Hyperthyroidism

Cases including events of hyperthyroidism are retrieved from the safety database for analysis if they contain an event PT within the 'Hyperthyroidism' SMQ (broad scope), i.e., any of the following MedDRA PTs:

| ANTI-THYROID ANTIBODY |
|---------------------------------|
| ANTI-THYROID ANTIBODY DECREASED |
| ANTI-THYROID ANTIBODY POSITIVE |
| ANTITHYROID ARTHRITIS SYNDROME |
| AUTOIMMUNE THYROID DISORDER |
| AUTOIMMUNE THYROIDITIS |

Status: Approved, Date: 2 May 2022

**BASEDOW'S DISEASE** 

BIOPSY THYROID GLAND ABNORMAL

BLOOD THYROID STIMULATING HORMONE ABNORMAL

BLOOD THYROID STIMULATING HORMONE DECREASED

BLOOD THYROID STIMULATING HORMONE INCREASED

BUTANOL-EXTRACTABLE IODINE DECREASED

BUTANOL-EXTRACTABLE IODINE INCREASED

CONGENITAL THYROID DISORDER

ENDOCRINE OPHTHALMOPATHY

**EUTHYROID SICK SYNDROME** 

**EXOPHTHALMOS** 

FREE THYROXINE INDEX ABNORMAL

FREE THYROXINE INDEX DECREASED

FREE THYROXINE INDEX INCREASED

GAMMA RADIATION THERAPY TO THYROID

**GOITRE** 

HASHIMOTO'S ENCEPHALOPATHY

**HASHITOXICOSIS** 

**HYPERTHYROIDISM** 

IMMUNE-MEDIATED HYPERTHYROIDISM

**IMMUNE-MEDIATED THYROIDITIS** 

INAPPROPRIATE THYROID STIMULATING HORMONE SECRETION

INFECTIOUS THYROIDITIS

IODINE UPTAKE ABNORMAL

IODINE UPTAKE DECREASED

IODINE UPTAKE INCREASED

MALIGNANT EXOPHTHALMOS

MARINE LENHART SYNDROME

ORBITAL DECOMPRESSION

PHOTON RADIATION THERAPY TO THYROID

POLYGLANDULAR AUTOIMMUNE SYNDROME TYPE II

POLYGLANDULAR AUTOIMMUNE SYNDROME TYPE III

PRIMARY HYPERTHYROIDISM

PROTEIN BOUND IODINE DECREASED

PROTEIN BOUND IODINE INCREASED

RADIOACTIVE IODINE THERAPY

RADIOTHERAPY TO THYROID

REVERSE TRI-IODOTHYRONINE DECREASED

REVERSE TRI-IODOTHYRONINE INCREASED

SECONDARY HYPERTHYROIDISM

SILENT THYROIDITIS

| THYREOSTATIC THERAPY |
|---------------------------------------------------|
| THYROGLOBULIN ABSENT |
| THYROGLOBULIN DECREASED |
| THYROGLOBULIN INCREASED |
| THYROGLOBULIN PRESENT |
| THYROID AUTOTRANSPLANTATION |
| THYROID DERMATOPATHY |
| THYROID DISORDER |
| THYROID DYSFUNCTION IN PREGNANCY |
| THYROID ELECTRON RADIATION THERAPY |
| THYROID FUNCTION TEST ABNORMAL |
| THYROID GLAND SCAN ABNORMAL |
| THYROID HEMIAGENESIS |
| THYROID HORMONE REPLACEMENT THERAPY |
| THYROID HORMONES INCREASED |
| THYROID OPERATION |
| THYROID PAIN |
| THYROID RELEASING HORMONE CHALLENGE TEST ABNORMAL |
| THYROID STIMULATING IMMUNOGLOBULIN INCREASED |
| THYROID THERAPY |
| THYROID TUBERCULOSIS |
| THYROIDECTOMY |
| THYROIDITIS |
| THYROIDITIS ACUTE |
| THYROIDITIS CHRONIC |
| THYROIDITIS FIBROUS CHRONIC |
| THYROIDITIS SUBACUTE |
| THYROTOXIC CARDIOMYOPATHY |
| THYROTOXIC CRISIS |
| THYROTOXIC MYOPATHY |
| THYROTOXIC PERIODIC PARALYSIS |
| THYROXIN BINDING GLOBULIN ABNORMAL |
| THYROXIN BINDING GLOBULIN DECREASED |
| THYROXIN BINDING GLOBULIN INCREASED |
| THYROXINE ABNORMAL |
| THYROXINE DECREASED |
| THYROXINE FREE ABNORMAL |
| THYROXINE FREE DECREASED |
| THYROXINE FREE INCREASED |
| THYROXINE INCREASED |
| THYROXINE THERAPY |

| TOXIC GOITRE |
|------------------------------------|
| TOXIC NODULAR GOITRE |
| TRI-IODOTHYRONINE ABNORMAL |
| TRI-IODOTHYRONINE DECREASED |
| TRI-IODOTHYRONINE FREE ABNORMAL |
| TRI-IODOTHYRONINE FREE DECREASED |
| TRI-IODOTHYRONINE FREE INCREASED |
| TRI-IODOTHYRONINE FREE NORMAL |
| TRI-IODOTHYRONINE INCREASED |
| TRI-IODOTHYRONINE UPTAKE ABNORMAL |
| TRI-IODOTHYRONINE UPTAKE DECREASED |
| TRI-IODOTHYRONINE UPTAKE INCREASED |
| ULTRASOUND THYROID ABNORMAL |
| X-RAY THERAPY TO THYROID |

## 1.5 Hypotension

"The case will be included in this subgroup if it contains an event with any of the following MedDRA Preferred Terms:

| BLOOD PRESSURE AMBULATORY DECREASED |
|-----------------------------------------------|
| BLOOD PRESSURE DECREASED |
| BLOOD PRESSURE DIASTOLIC DECREASED |
| BLOOD PRESSURE IMMEASURABLE |
| BLOOD PRESSURE ORTHOSTATIC DECREASED |
| BLOOD PRESSURE SYSTOLIC DECREASED |
| BLOOD PRESSURE SYSTOLIC INSPIRATORY DECREASED |
| CT HYPOTENSION COMPLEX |
| DIALYSIS HYPOTENSION |
| DIASTOLIC HYPOTENSION |
| HYPOTENSION |
| HYPOTENSIVE CRISIS |
| MEAN ARTERIAL PRESSURE DECREASED |
| NEONATAL HYPOTENSION |
| ORTHOSTATIC HYPOTENSION |
| POST PROCEDURAL HYPOTENSION |
| PROCEDURAL HYPOTENSION |

# 1.6 Light-dependent non-melanoma skin malignancies

Cases including events denoting non-melanoma skin malignancies are retrieved from the safety database for analysis if they contain an event PT within the MedDRA High Level Term 'Skin neoplasms malignant and unspecified (excl. melanoma)', or if they contain the MedDRA PT 'Squamous cell carcinoma', i.e., any of the following MedDRA PTs:

ATYPICAL FIBROXANTHOMA

BASAL CELL CARCINOMA BASAL CELL CARCINOMA METASTATIC BASAL CELL NAEVUS SYNDROME BASOSQUAMOUS CARCINOMA OF SKIN **BOWEN'S DISEASE** CARCINOMA IN SITU OF SKIN DYSPLASTIC NAEVUS SYNDROME ECCRINE CARCINOMA EPIDERMAL NAEVUS SYNDROME EXTRAMAMMARY PAGET'S DISEASE HIDRADENOCARCINOMA KERATOACANTHOMA MALIGNANT SWEAT GLAND NEOPLASM MARJOLIN'S ULCER MASTOCYTOMA NEOPLASM SKIN NEUROENDOCRINE CARCINOMA OF THE SKIN PILOMATRIX CARCINOMA POROCARCINOMA SEBACEOUS CARCINOMA SKIN ANGIOSARCOMA SKIN CANCER SKIN CANCER METASTATIC SKIN NEOPLASM BLEEDING SKIN SQUAMOUS CELL CARCINOMA METASTATIC SKIN SQUAMOUS CELL CARCINOMA RECURRENT SQUAMOUS CELL CARCINOMA

# 1.7 Major adverse cardiovascular events

SQUAMOUS CELL CARCINOMA OF SKIN

TRICHOBLASTIC CARCINOMA

Cases including major adverse cardiovascular events (MACE) are retrieved from the safety database for analysis if they contain an event PT within any of the following MedDRA SMQs: 'Conditions associated with central nervous system haemorrhages and cerebrovascular accidents' (broad scope), 'Haemorrhagic central nervous system vascular conditions' (narrow scope), 'Ischaemic central nervous system vascular conditions' (narrow scope), or 'Myocardial infarction' (narrow scope), or an event with any of the following MedDRA PTs: 'Cardiac arrest', 'Cardiac death', 'Cardio-respiratory arrest', 'Coronary artery disease', 'Coronary artery insufficiency', 'Coronary vein stenosis', 'Myocardial ischaemia', 'Pseudostroke', 'Sudden cardiac death', and 'Sudden death', i.e., any of the following MedDRA PTs:

ACUTE CARDIAC EVENT
ACUTE CORONARY SYNDROME

CONFIDENTIAL – FOIA Exemptions Apply in U.S.

| ACUTE MYOCARDIAL INFARCTION |
|-------------------------------------------|
| AGNOSIA |
| AMAUROSIS FUGAX |
| ANGINA UNSTABLE |
| ANGIOGRAM CEREBRAL ABNORMAL |
| APHASIA |
| BALINT'S SYNDROME |
| BASAL GANGLIA HAEMATOMA |
| BASAL GANGLIA HAEMORRHAGE |
| BASAL GANGLIA INFARCTION |
| BASAL GANGLIA STROKE |
| BASILAR ARTERY ANEURYSM |
| BASILAR ARTERY OCCLUSION |
| BASILAR ARTERY PERFORATION |
| BASILAR ARTERY STENOSIS |
| BASILAR ARTERY THROMBOSIS |
| BENEDIKT'S SYNDROME |
| BLOOD CREATINE PHOSPHOKINASE MB ABNORMAL |
| BLOOD CREATINE PHOSPHOKINASE MB INCREASED |
| BRACHIOCEPHALIC ARTERIOSCLEROSIS |
| BRACHIOCEPHALIC ARTERY OCCLUSION |
| BRACHIOCEPHALIC ARTERY STENOSIS |
| BRAIN HYPOXIA |
| BRAIN INJURY |
| BRAIN STEM EMBOLISM |
| BRAIN STEM HAEMATOMA |
| BRAIN STEM HAEMORRHAGE |
| BRAIN STEM INFARCTION |
| BRAIN STEM ISCHAEMIA |
| BRAIN STEM MICROHAEMORRHAGE |
| BRAIN STEM STROKE |
| BRAIN STEM THROMBOSIS |
| BRAIN STENT INSERTION |
| CADASIL |
| CAPSULAR WARNING SYNDROME |
| CARASIL SYNDROME |
| CARDIAC ARREST |
| CARDIAC DEATH |
| CARDIO-RESPIRATORY ARREST |
| CAROTID ANEURYSM RUPTURE |
| CAROTID ANGIOPLASTY |

| CAROTID ARTERIAL EMBOLUS |
|--------------------------------------------------|
| CAROTID ARTERIOSCLEROSIS |
| CAROTID ARTERY ANEURYSM |
| CAROTID ARTERY BYPASS |
| CAROTID ARTERY DISEASE |
| CAROTID ARTERY DISSECTION |
| CAROTID ARTERY INSUFFICIENCY |
| CAROTID ARTERY OCCLUSION |
| CAROTID ARTERY PERFORATION |
| CAROTID ARTERY RESTENOSIS |
| CAROTID ARTERY STENOSIS |
| CAROTID ARTERY STENT INSERTION |
| CAROTID ARTERY STENT REMOVAL |
| CAROTID ARTERY THROMBOSIS |
| CAROTID ENDARTERECTOMY |
| CAROTID REVASCULARISATION |
| CENTRAL NERVOUS SYSTEM HAEMORRHAGE |
| CENTRAL PAIN SYNDROME |
| CEREBELLAR ARTERY OCCLUSION |
| CEREBELLAR ARTERY THROMBOSIS |
| CEREBELLAR ATHEROSCLEROSIS |
| CEREBELLAR EMBOLISM |
| CEREBELLAR HAEMATOMA |
| CEREBELLAR HAEMORRHAGE |
| CEREBELLAR INFARCTION |
| CEREBELLAR ISCHAEMIA |
| CEREBELLAR MICROHAEMORRHAGE |
| CEREBELLAR STROKE |
| CEREBRAL ANEURYSM PERFORATION |
| CEREBRAL ANEURYSM RUPTURED SYPHILITIC |
| CEREBRAL ARTERIOSCLEROSIS |
| CEREBRAL ARTERIOVENOUS MALFORMATION HAEMORRHAGIC |
| CEREBRAL ARTERY EMBOLISM |
| CEREBRAL ARTERY OCCLUSION |
| CEREBRAL ARTERY PERFORATION |
| CEREBRAL ARTERY RESTENOSIS |
| CEREBRAL ARTERY STENOSIS |
| CEREBRAL ARTERY STENT INSERTION |
| CEREBRAL ARTERY THROMBOSIS |
| CEREBRAL CAVERNOUS MALFORMATION |
| CEREBRAL CYST HAEMORRHAGE |

| CEREBRAL ENDOVASCULAR ANEURYSM REPAIR |
|-----------------------------------------|
| CEREBRAL GAS EMBOLISM |
| CEREBRAL HAEMATOMA |
| CEREBRAL HAEMORRHAGE |
| CEREBRAL HAEMORRHAGE FOETAL |
| CEREBRAL HAEMORRHAGE NEONATAL |
| CEREBRAL HAEMOSIDERIN DEPOSITION |
| CEREBRAL INFARCTION |
| CEREBRAL INFARCTION FOETAL |
| CEREBRAL ISCHAEMIA |
| CEREBRAL MICROEMBOLISM |
| CEREBRAL MICROHAEMORRHAGE |
| CEREBRAL MICROINFARCTION |
| CEREBRAL REPERFUSION INJURY |
| CEREBRAL REVASCULARISATION |
| CEREBRAL SEPTIC INFARCT |
| CEREBRAL SMALL VESSEL ISCHAEMIC DISEASE |
| CEREBRAL THROMBOSIS |
| CEREBRAL VASCULAR OCCLUSION |
| CEREBRAL VASOCONSTRICTION |
| CEREBRAL VENOUS THROMBOSIS |
| CEREBRAL VENTRICULAR RUPTURE |
| CEREBROVASCULAR ACCIDENT |
| CEREBROVASCULAR ACCIDENT PROPHYLAXIS |
| CEREBROVASCULAR DISORDER |
| CEREBROVASCULAR INSUFFICIENCY |
| CEREBROVASCULAR PSEUDOANEURYSM |
| CEREBROVASCULAR STENOSIS |
| CHARCOT-BOUCHARD MICROANEURYSMS |
| CLAUDE'S SYNDROME |
| CONGENITAL HEMIPARESIS |
| CORONARY ARTERY DISEASE |
| CORONARY ARTERY EMBOLISM |
| CORONARY ARTERY INSUFFICIENCY |
| CORONARY ARTERY OCCLUSION |
| CORONARY ARTERY REOCCLUSION |
| CORONARY ARTERY THROMBOSIS |
| CORONARY BYPASS THROMBOSIS |
| CORONARY VASCULAR GRAFT OCCLUSION |
| CORONARY VEIN STENOSIS |
| CSF BILIRUBIN POSITIVE |

CSF RED BLOOD CELL COUNT POSITIVE DELAYED ISCHAEMIC NEUROLOGICAL DEFICIT DIPLEGIA **DYSARTHRIA** EMBOLIC CEREBELLAR INFARCTION EMBOLIC CEREBRAL INFARCTION EMBOLIC STROKE EPIDURAL HAEMORRHAGE EXTRA-AXIAL HAEMORRHAGE EXTRADURAL HAEMATOMA EXTRADURAL HAEMATOMA EVACUATION EXTRAISCHAEMIC CEREBRAL HAEMATOMA FOVILLE SYNDROME HAEMORRHAGE INTRACRANIAL HAEMORRHAGIC CEREBRAL INFARCTION HAEMORRHAGIC STROKE HAEMORRHAGIC TRANSFORMATION STROKE HEMIANAESTHESIA **HEMIASOMATOGNOSIA HEMIATAXIA HEMIDYSAESTHESIA HEMIHYPERAESTHESIA HEMIPARAESTHESIA HEMIPARESIS** HEMIPLEGIA HUNT AND HESS SCALE HYPOXIC-ISCHAEMIC ENCEPHALOPATHY INNER EAR INFARCTION INTERNAL CAPSULE INFARCTION INTERNAL CAROTID ARTERY DEFORMITY INTRA-CEREBRAL ANEURYSM OPERATION INTRACEREBRAL HAEMATOMA EVACUATION INTRACRANIAL ANEURYSM INTRACRANIAL ARTERY DISSECTION INTRACRANIAL HAEMATOMA INTRACRANIAL TUMOUR HAEMORRHAGE INTRAVENTRICULAR HAEMORRHAGE INTRAVENTRICULAR HAEMORRHAGE NEONATAL ISCHAEMIC CEREBRAL INFARCTION ISCHAEMIC STROKE **KOUNIS SYNDROME** 

CONFIDENTIAL – FOIA Exemptions Apply in U.S.

LACUNAR INFARCTION LACUNAR STROKE LATERAL MEDULLARY SYNDROME LATEROPULSION MENINGORRHAGIA MIGRAINOUS INFARCTION MILLARD-GUBLER SYNDROME MODIFIED RANKIN SCORE DECREASED MODIFIED RANKIN SCORE INCREASED **MONOPARESIS MONOPLEGIA** MOYAMOYA DISEASE MYOCARDIAL INFARCTION MYOCARDIAL ISCHAEMIA MYOCARDIAL NECROSIS MYOCARDIAL REPERFUSION INJURY MYOCARDIAL STUNNING NIH STROKE SCALE ABNORMAL NIH STROKE SCALE SCORE DECREASED NIH STROKE SCALE SCORE INCREASED PAPILLARY MUSCLE INFARCTION **PARALYSIS PARAPARESIS PARAPLEGIA PARESIS** PERINATAL STROKE PERIPROCEDURAL MYOCARDIAL INFARCTION PERIVENTRICULAR HAEMORRHAGE NEONATAL PITUITARY APOPLEXY PITUITARY HAEMORRHAGE POST CARDIAC ARREST SYNDROME POST PROCEDURAL MYOCARDIAL INFARCTION POST PROCEDURAL STROKE POST STROKE DEPRESSION POSTHAEMORRHAGIC HYDROCEPHALUS POSTINFARCTION ANGINA PRECEREBRAL ARTERIOSCLEROSIS PRECEREBRAL ARTERY EMBOLISM PRECEREBRAL ARTERY OCCLUSION PRECEREBRAL ARTERY THROMBOSIS PSEUDOSTROKE

CONFIDENTIAL – FOIA Exemptions Apply in U.S.

PUTAMEN HAEMORRHAGE **QUADRIPARESIS QUADRIPLEGIA** REVERSIBLE CEREBRAL VASOCONSTRICTION SYNDROME REVERSIBLE ISCHAEMIC NEUROLOGICAL DEFICIT RIGHT HEMISPHERE DEFICIT SYNDROME RUPTURED CEREBRAL ANEURYSM SILENT MYOCARDIAL INFARCTION SPINAL ARTERY EMBOLISM SPINAL ARTERY THROMBOSIS SPINAL CORD HAEMATOMA SPINAL CORD HAEMORRHAGE SPINAL CORD INFARCTION SPINAL CORD ISCHAEMIA SPINAL EPIDURAL HAEMATOMA SPINAL EPIDURAL HAEMORRHAGE SPINAL STROKE SPINAL SUBARACHNOID HAEMORRHAGE SPINAL SUBDURAL HAEMATOMA SPINAL SUBDURAL HAEMORRHAGE STROKE IN EVOLUTION SUBARACHNOID HAEMATOMA SUBARACHNOID HAEMORRHAGE SUBARACHNOID HAEMORRHAGE NEONATAL SUBCLAVIAN STEAL SYNDROME SUBDURAL HAEMATOMA SUBDURAL HAEMATOMA EVACUATION SUBDURAL HAEMORRHAGE SUBDURAL HAEMORRHAGE NEONATAL SUDDEN CARDIAC DEATH SUDDEN DEATH SUPERFICIAL SIDEROSIS OF CENTRAL NERVOUS SYSTEM THALAMIC INFARCTION THALAMUS HAEMORRHAGE THROMBOTIC CEREBRAL INFARCTION THROMBOTIC STROKE TRANSIENT ISCHAEMIC ATTACK TROPONIN I INCREASED TROPONIN INCREASED TROPONIN T INCREASED

CONFIDENTIAL – FOIA Exemptions Apply in U.S.

VASCULAR ENCEPHALOPATHY

VASCULAR STENT OCCLUSION

VASCULAR STENT STENOSIS

VEIN OF GALEN ANEURYSMAL MALFORMATION

VERTEBRAL ARTERY ANEURYSM

VERTEBRAL ARTERY ARTERIOSCLEROSIS

VERTEBRAL ARTERY DISSECTION

VERTEBRAL ARTERY OCCLUSION

VERTEBRAL ARTERY PERFORATION

VERTEBRAL ARTERY STENOSIS

VERTEBRAL ARTERY THROMBOSIS

VERTEBROBASILAR INSUFFICIENCY

VERTEBROBASILAR STROKE

VISUAL AGNOSIA

VISUAL MIDLINE SHIFT SYNDROME

WEBER'S SYNDROME

## 1.8 Medication errors

Cases with events of medication errors are retrieved from the safety database for analysis if they contain an event PT within the 'Medication errors' SMQ (narrow scope), i.e., any of the following MedDRA PTs:

| ACCIDENTAL DEVICE INGESTION |
|--------------------------------------------------------------------|
| ACCIDENTAL DEVICE INGESTION BY A CHILD |
| ACCIDENTAL EXPOSURE TO PRODUCT |
| ACCIDENTAL EXPOSURE TO PRODUCT BY CHILD |
| ACCIDENTAL EXPOSURE TO PRODUCT PACKAGING |
| ACCIDENTAL EXPOSURE TO PRODUCT PACKAGING BY CHILD |
| ACCIDENTAL OVERDOSE |
| ACCIDENTAL POISONING |
| ACCIDENTAL UNDERDOSE |
| ACCIDENTAL USE OF PLACEBO |
| BOOSTER DOSE MISSED |
| CIRCUMSTANCE OR INFORMATION CAPABLE OF LEADING TO DEVICE USE ERROR |
| CIRCUMSTANCE OR INFORMATION CAPABLE OF LEADING TO MEDICATION ERROR |
| CONTRAINDICATED DEVICE USED |
| CONTRAINDICATED PRODUCT ADMINISTERED |
| CONTRAINDICATED PRODUCT PRESCRIBED |
| DEPRESCRIBING ERROR |
| DEVICE DISPENSING ERROR |
| DEVICE MONITORING PROCEDURE NOT PERFORMED |
| DEVICE PROGRAMMING ERROR |
| DEVICE USE CONFUSION |

CONFIDENTIAL – FOIA Exemptions Apply in U.S.

DEVICE USE ERROR
DISCONTINUED PRODUCT ADMINISTERED

DOCUMENTED HYPERSENSITIVITY TO ADMINISTERED PRODUCT

DOSE CALCULATION ERROR

DRUG ADMINISTERED IN WRONG DEVICE

DRUG DISPENSED TO WRONG PATIENT

DRUG DOSE OMISSION BY DEVICE

DRUG DOSE TITRATION NOT PERFORMED

DRUG MONITORING PROCEDURE INCORRECTLY PERFORMED

DRUG MONITORING PROCEDURE NOT PERFORMED

DRUG TITRATION ERROR

**DUPLICATE THERAPY ERROR** 

EXPIRED DEVICE USED

EXPIRED PRODUCT ADMINISTERED

EXPOSURE VIA DIRECT CONTACT

EXPOSURE VIA EYE CONTACT

EXPOSURE VIA SKIN CONTACT

EXTRA DOSE ADMINISTERED

FAILURE OF CHILD RESISTANT PRODUCT CLOSURE

FAILURE TO SUSPEND MEDICATION

INADEQUATE ASEPTIC TECHNIQUE IN USE OF PRODUCT

INAPPROPRIATE SCHEDULE OF PRODUCT ADMINISTRATION

INAPPROPRIATE SCHEDULE OF PRODUCT DISCONTINUATION

INCOMPLETE COURSE OF VACCINATION

INCORRECT DISPOSAL OF PRODUCT

INCORRECT DOSAGE ADMINISTERED

INCORRECT DOSE ADMINISTERED

INCORRECT DOSE ADMINISTERED BY DEVICE

INCORRECT DOSE ADMINISTERED BY PRODUCT

INCORRECT DRUG ADMINISTRATION RATE

INCORRECT PRODUCT ADMINISTRATION DURATION

INCORRECT PRODUCT DOSAGE FORM ADMINISTERED

INCORRECT PRODUCT FORMULATION ADMINISTERED

INCORRECT ROUTE OF PRODUCT ADMINISTRATION

INTERCEPTED ACCIDENTAL EXPOSURE TO PRODUCT BY CHILD

INTERCEPTED MEDICATION ERROR

INTERCEPTED PRODUCT ADMINISTRATION ERROR

INTERCEPTED PRODUCT DISPENSING ERROR

INTERCEPTED PRODUCT MONITORING ERROR

INTERCEPTED PRODUCT PREPARATION ERROR

INTERCEPTED PRODUCT PRESCRIBING ERROR

INTERCEPTED PRODUCT SELECTION ERROR INTERCEPTED PRODUCT STORAGE ERROR INTERCEPTED WRONG PATIENT SELECTED LABELLED DRUG-DISEASE INTERACTION MEDICATION ERROR LABELLED DRUG-DRUG INTERACTION MEDICATION ERROR LABELLED DRUG-FOOD INTERACTION MEDICATION ERROR LACK OF ADMINISTRATION SITE ROTATION LACK OF APPLICATION SITE ROTATION LACK OF INFUSION SITE ROTATION LACK OF INJECTION SITE ROTATION LACK OF VACCINATION SITE ROTATION MEDICAL DEVICE MONITORING ERROR MEDICATION ERROR MULTIPLE USE OF SINGLE-USE PRODUCT PARAVENOUS DRUG ADMINISTRATION PRODUCT ADMINISTERED AT INAPPROPRIATE SITE PRODUCT ADMINISTERED BY WRONG PERSON PRODUCT ADMINISTERED TO PATIENT OF INAPPROPRIATE AGE PRODUCT ADMINISTRATION ERROR PRODUCT APPEARANCE CONFUSION PRODUCT BARCODE ISSUE PRODUCT CONFUSION PRODUCT DESIGN CONFUSION PRODUCT DISPENSING ERROR PRODUCT DOSAGE FORM CONFUSION PRODUCT DOSE OMISSION IN ERROR PRODUCT LABEL CONFUSION PRODUCT MONITORING ERROR PRODUCT NAME CONFUSION PRODUCT PACKAGING CONFUSION PRODUCT PREPARATION ERROR PRODUCT PRESCRIBING ERROR PRODUCT SELECTION ERROR PRODUCT STORAGE ERROR PRODUCT SUBSTITUTION ERROR RECALLED PRODUCT ADMINISTERED SINGLE COMPONENT OF A TWO-COMPONENT PRODUCT ADMINISTERED THERAPEUTIC DRUG MONITORING ANALYSIS INCORRECTLY PERFORMED THERAPEUTIC DRUG MONITORING ANALYSIS NOT PERFORMED TRANSCRIPTION MEDICATION ERROR

Status: Approved, Date: 2 May 2022

TRANSFUSION WITH INCOMPATIBLE BLOOD

UNINTENTIONAL USE FOR UNAPPROVED INDICATION VACCINATION ERROR WRONG DEVICE USED WRONG DOSAGE FORM WRONG DOSAGE FORMULATION WRONG DOSE WRONG DRUG WRONG PATIENT WRONG PATIENT RECEIVED PRODUCT WRONG PRODUCT ADMINISTERED WRONG PRODUCT PROCURED WRONG PRODUCT STORED WRONG RATE WRONG ROUTE WRONG SCHEDULE WRONG STRENGTH WRONG TECHNIQUE IN DEVICE USAGE PROCESS WRONG TECHNIQUE IN PRODUCT USAGE PROCESS

# 1.9 Ophthalmological effects associated with retinal vascular system

Cases describing ophthalmological effects associated with the retinal vascular system are retrieved from the safety database for analysis if they contain an event PT within the 'Retinal disorders' SMQ (broad scope), i.e., any of the following MedDRA PTs:

| ACQUIRED PIGMENTED RETINOPATHY |
|--------------------------------------|
| ACUTE MACULAR OUTER RETINOPATHY |
| ACUTE ZONAL OCCULT OUTER RETINOPATHY |
| AGE-RELATED MACULAR DEGENERATION |
| AIDS RETINOPATHY |
| AMAUROSIS FUGAX |
| ANGIOGRAM RETINA ABNORMAL |
| ARTERIOSCLEROTIC RETINOPATHY |
| AUTOIMMUNE EYE DISORDER |
| AUTOIMMUNE RETINOPATHY |
| BENIGN NEOPLASM OF RETINA |
| BIOPSY RETINA ABNORMAL |
| BIRDSHOT CHORIORETINOPATHY |
| BLINDNESS |
| BLINDNESS TRANSIENT |
| BLINDNESS UNILATERAL |
| CENTRAL VISION LOSS |
| CHOLESTEROLOSIS BULBI |

CONFIDENTIAL – FOIA Exemptions Apply in U.S.

A COLUDED DICMENTED DETINODATIV

Statistical Analysis Plan AC-065A203; Amendment 7 CHORIORETINAL ATROPHY CHORIORETINAL DISORDER CHORIORETINAL SCAR **CHORIORETINITIS** CHORIORETINOPATHY CHOROIDAL OSTEOMA **CHROMATOPSIA** CILIARY BODY MELANOMA **COLOUR BLINDNESS** COLOUR BLINDNESS ACQUIRED COLOUR VISION TESTS ABNORMAL COLOUR VISION TESTS ABNORMAL BLUE-YELLOW COLOUR VISION TESTS ABNORMAL RED-GREEN COMMOTIO RETINAE CYSTOID MACULAR OEDEMA **DELAYED LIGHT ADAPTATION** DETACHMENT OF MACULAR RETINAL PIGMENT EPITHELIUM DETACHMENT OF RETINAL PIGMENT EPITHELIUM DIABETIC RETINAL OEDEMA DIABETIC RETINOPATHY DIFFUSE UVEAL MELANOCYTIC PROLIFERATION DISRUPTION OF THE PHOTORECEPTOR INNER SEGMENT-OUTER SEGMENT DRY AGE-RELATED MACULAR DEGENERATION DYSCHROMATOPSIA EXTRAOCULAR RETINOBLASTOMA **EXUDATIVE RETINOPATHY** EYE DISORDER EYE HAEMATOMA EYE HAEMORRHAGE **EYE INFARCTION** EYE NAEVUS EYE OPACITY FLUORESCENCE ANGIOGRAM ABNORMAL FOVEAL DEGENERATION FOVEAL REFLEX ABNORMAL FUNDOSCOPY ABNORMAL HAEMORRHAGIC OCCLUSIVE RETINAL VASCULITIS

CONFIDENTIAL - FOIA Exemptions Apply in U.S.

HYPERTENSIVE CEREBROVASCULAR DISEASE

62

HYPOTONY MACULOPATHY IMMUNE RECOVERY UVEITIS

HYPERAESTHESIA EYE

Statistical Analysis Plan AC-065A203; Amendment 7 **IMMUNE-MEDIATED UVEITIS** INTERNAL LIMITING MEMBRANE PEELING INTRA-OCULAR INJECTION COMPLICATION INTRAOCULAR HAEMATOMA INTRAVITREAL IMPLANT **IRVAN SYNDROME** LEUKAEMIC RETINOPATHY LEUKOCORIA LIPAEMIA RETINALIS LOW LUMINANCE BEST-CORRECTED VISUAL ACUITY DECREASED MACULAR CYST MACULAR DEGENERATION MACULAR DETACHMENT **MACULAR FIBROSIS** MACULAR HOLE MACULAR ISCHAEMIA MACULAR OEDEMA MACULAR OPACITY **MACULAR PIGMENTATION** MACULAR PSEUDOHOLE MACULAR REFLEX ABNORMAL MACULAR RUPTURE MACULAR SCAR MACULAR TELANGIECTASIA MACULAR THICKENING **MACULOPATHY** MALIGNANT NEOPLASM OF RETINA METAMORPHOPSIA MYOPIC CHORIORETINAL DEGENERATION MYOPIC TRACTION MACULOPATHY NECROTISING RETINITIS NEOVASCULAR AGE-RELATED MACULAR DEGENERATION NEUROPATHY, ATAXIA, RETINITIS PIGMENTOSA SYNDROME NON-PROLIFERATIVE RETINOPATHY NONINFECTIVE CHORIORETINITIS

NONINFECTIVE RETINITIS

OCULAR ISCHAEMIC SYNDROME

OCULAR LYMPHOMA

OCULAR STEM CELL TRANSPLANT

OPHTHALMIC ARTERY THROMBOSIS

OPHTHALMIC VEIN THROMBOSIS

OPTIC DISC TRACTION SYNDROME OPTICAL COHERENCE TOMOGRAPHY ABNORMAL ORBITAL HAEMATOMA ORBITAL HAEMORRHAGE PARANEOPLASTIC RETINOPATHY PARS PLANA CYST PATHOLOGIC MYOPIA PERIPAPILLARY PIGMENTATION PHOTOPHOBIA **PHOTOPSIA** POST THROMBOTIC RETINOPATHY PUPILLARY LIGHT REFLEX TESTS ABNORMAL PURTSCHER RETINOPATHY RADIATION RETINOPATHY RED REFLEX ABNORMAL **RETINAL ANEURYSM** RETINAL ANEURYSM RUPTURE RETINAL ARTERIOVENOUS MALFORMATION RETINAL ARTERY EMBOLISM RETINAL ARTERY OCCLUSION RETINAL ARTERY SPASM RETINAL ARTERY STENOSIS RETINAL ARTERY THROMBOSIS RETINAL COLLATERAL VESSELS RETINAL COLOBOMA RETINAL CRYOABLATION **RETINAL CYST** RETINAL CYST EXCISION RETINAL DEGENERATION RETINAL DEPIGMENTATION RETINAL DEPOSITS RETINAL DETACHMENT RETINAL DISORDER RETINAL DRUSEN RETINAL DYSTROPHY RETINAL EXUDATES **RETINAL FIBROSIS** RETINAL FOVEA DISORDER RETINAL FUNCTION TEST ABNORMAL RETINAL HAEMORRHAGE RETINAL IMPLANT

CONFIDENTIAL – FOIA Exemptions Apply in U.S.

| RETINAL INFARCTION |
|---------------------------------|
| RETINAL INFILTRATES |
| RETINAL INJURY |
| RETINAL ISCHAEMIA |
| RETINAL LASER COAGULATION |
| RETINAL MELANOCYTOMA |
| RETINAL MELANOMA |
| RETINAL MIGRAINE |
| RETINAL NEOPLASM |
| RETINAL NEOVASCULARISATION |
| RETINAL OCCLUSIVE VASCULITIS |
| RETINAL OEDEMA |
| RETINAL OPERATION |
| RETINAL PALLOR |
| RETINAL PERIVASCULAR SHEATHING |
| RETINAL PHOTOTOXICITY |
| RETINAL PIGMENT EPITHELIAL TEAR |
| RETINAL PIGMENT EPITHELIOPATHY |
| RETINAL PIGMENTATION |
| RETINAL SCAR |
| RETINAL TEAR |
| RETINAL TELANGIECTASIA |
| RETINAL THICKENING |
| RETINAL TOXICITY |
| RETINAL TRANSPLANT |
| RETINAL TUMOUR EXCISION |
| RETINAL VASCULAR DISORDER |
| RETINAL VASCULAR OCCLUSION |
| RETINAL VASCULAR THROMBOSIS |
| RETINAL VASCULITIS |
| RETINAL VEIN OCCLUSION |
| RETINAL VEIN THROMBOSIS |
| RETINAL VEIN VARICES |
| RETINAL VESSEL AVULSION |
| RETINAL WHITE WITHOUT PRESSURE |
| RETINITIS |
| RETINITIS PIGMENTOSA |
| RETINOBLASTOMA |
| RETINOGRAM ABNORMAL |
| RETINOPATHY |
| RETINOPATHY HAEMORRHAGIC |

RETINOPATHY HYPERTENSIVE
RETINOPATHY HYPERVISCOSITY

RETINOPATHY OF PREMATURITY

RETINOPATHY PROLIFERATIVE

RETINOPATHY SICKLE CELL

RETINOPATHY SOLAR

RETINOPEXY

RETINOSCHISIS

RHEGMATOGENOUS RETINAL DETACHMENT

SCINTILLATING SCOTOMA

SCLERAL BUCKLING SURGERY

**SCLEROTOMY** 

SEROUS RETINAL DETACHMENT

SEROUS RETINOPATHY

**SERPIGINOUS CHOROIDITIS** 

SUBRETINAL FIBROSIS

SUBRETINAL FLUID

SUBRETINAL HAEMATOMA

SUBRETINAL HYPERREFLECTIVE EXUDATION

SUSAC'S SYNDROME

**TESSELLATED FUNDUS** 

TRACTIONAL RETINAL DETACHMENT

TRANSPUPILLARY THERMOTHERAPY

**TUNNEL VISION** 

UVEAL MELANOMA

VASCULAR ENDOTHELIAL GROWTH FACTOR OVEREXPRESSION

VENOUS STASIS RETINOPATHY

**VISION BLURRED** 

VISUAL ACUITY REDUCED

VISUAL ACUITY TESTS ABNORMAL

VISUAL FIELD DEFECT

VISUAL FIELD TESTS ABNORMAL

VISUAL IMPAIRMENT

VITREAL CELLS

VITRECTOMY

VITREOMACULAR INTERFACE ABNORMAL

VITREORETINAL TRACTION SYNDROME

VITREOUS ADHESIONS

VITREOUS DETACHMENT

VITREOUS DISORDER

VITREOUS FLOATERS

| VITREOUS HAEMATOMA |
|------------------------------|
| VITREOUS HAEMORRHAGE |
| VITREOUS HAZE |
| VITRITIS |
| VOGT-KOYANAGI-HARADA DISEASE |
| XANTHOPSIA |

## 1.10 Pregnancy

Cases referring to pregnancy are retrieved from the safety database for analysis if they meet any of the following conditions:

The case contains an event with a primary MedDRA System Organ Class containing the text: 'pregnancy' (but excluding the MedDRA PTs: 'Pregnancy test urine negative', 'Pregnancy test negative', or 'Pregnancy test false positive'),

OR

It contains an event with a MedDRA primary HLT or PT containing the following text: 'abortion', or 'pregnancy' (but excluding the PT 'Woman of childbearing potential').

OR

It contains an event with any of the following MedDRA PTs: 'Maternal drugs affecting foetus', 'Miscarriage of partner', or 'Paternal drugs affecting foetus', i.e., any of the following MedDRA PTs:

| ABNORMAL CORD INSERTION |
|-----------------------------------------|
| ABNORMAL LABOUR |
| ABNORMAL LABOUR AFFECTING FOETUS |
| ABNORMAL PRODUCT OF CONCEPTION |
| ABORTED PREGNANCY |
| ABORTION |
| ABORTION COMPLETE |
| ABORTION COMPLETE COMPLICATED |
| ABORTION COMPLICATED |
| ABORTION EARLY |
| ABORTION INCOMPLETE |
| ABORTION INCOMPLETE COMPLICATED |
| ABORTION INDUCED |
| ABORTION INDUCED COMPLETE |
| ABORTION INDUCED COMPLETE COMPLICATED |
| ABORTION INDUCED COMPLICATED |
| ABORTION INDUCED INCOMPLETE |
| ABORTION INDUCED INCOMPLETE COMPLICATED |
| ABORTION INFECTED |
| ABORTION LATE |
| ABORTION MISSED |

CONFIDENTIAL – FOIA Exemptions Apply in U.S.

Statistical Analysis Plan AC-065A203; Amendment 7 ABORTION OF ECTOPIC PREGNANCY ABORTION SPONTANEOUS ABORTION SPONTANEOUS COMPLETE ABORTION SPONTANEOUS COMPLETE COMPLICATED ABORTION SPONTANEOUS COMPLICATED ABORTION SPONTANEOUS INCOMPLETE ABORTION SPONTANEOUS INCOMPLETE COMPLICATED ABORTION THREATENED **ACUTE FATTY LIVER OF PREGNANCY** ADRENOCORTICAL INSUFFICIENCY NEONATAL AFTERBIRTH PAIN **AMNIORRHEXIS AMNIORRHOEA** AMNIOTIC CAVITY DISORDER ANAEMIA OF PREGNANCY ANAESTHETIC COMPLICATION NEONATAL ANAPHYLACTOID SYNDROME OF PREGNANCY ANEMBRYONIC GESTATION ARRESTED LABOUR ASYNCLITIC PRESENTATION **BACTERIURIA IN PREGNANCY BIOCHEMICAL PREGNANCY BIRTH TRAUMA BIRTH WEIGHT NORMAL BOTTLE FEEDING** BREAST ENGORGEMENT IN NEWBORN **BREAST FEEDING BREECH DELIVERY BREECH PRESENTATION BROW PRESENTATION** CAPUT SUCCEDANEUM **CEPHALHAEMATOMA** 

CEPHALO-PELVIC DISPROPORTION

**CERVICAL DILATATION** 

CERVICAL INCOMPETENCE

CERVIX DYSTOCIA

CHILD BORN TO UNMARRIED PARENTS

CHOLESTASIS OF PREGNANCY

CHORIOAMNIOTIC SEPARATION

CHRONIC VILLITIS OF UNKNOWN ETIOLOGY

COMPLICATION OF DELIVERY

COMPLICATION OF PREGNANCY

CRANIAL NERVE INJURY SECONDARY TO BIRTH TRAUMA

DECIDUAL CAST

**DELAYED DELIVERY** 

**DELIVERY** 

DELIVERY OUTSIDE HEALTH FACILITY

DIABETES COMPLICATING PREGNANCY

DISCORDANT TWIN

DRUG EXPOSURE BEFORE PREGNANCY

**ECLAMPSIA** 

**ECTOPIC PREGNANCY** 

ECTOPIC PREGNANCY TERMINATION

ECTOPIC PREGNANCY UNDER HORMONAL CONTRACEPTION

ECTOPIC PREGNANCY WITH CONTRACEPTIVE DEVICE

**ELDERLY PRIMIGRAVIDA** 

**EXPOSURE DURING PREGNANCY** 

EXPOSURE VIA BREAST MILK

EXPOSURE VIA FATHER

**FACE PRESENTATION** 

FACIAL NERVE INJURY DUE TO BIRTH TRAUMA

FAILED INDUCTION OF LABOUR

FAILED TRIAL OF LABOUR

FALSE LABOUR

FALSE NEGATIVE PREGNANCY TEST

FEAR OF PREGNANCY

FIRST TRIMESTER PREGNANCY

FOETAL ACIDOSIS

FOETAL ARM PROLAPSE

FOETAL CARDIAC DISORDER

FOETAL COMPARTMENT FLUID COLLECTION

FOETAL DAMAGE

FOETAL DEATH

FOETAL DISORDER

FOETAL DISTRESS SYNDROME

FOETAL DYSTOCIA

FOETAL EXPOSURE DURING DELIVERY

FOETAL EXPOSURE DURING PREGNANCY

FOETAL EXPOSURE TIMING UNSPECIFIED

FOETAL GROWTH ABNORMALITY

FOETAL GROWTH RESTRICTION

FOETAL HYPOKINESIA

FOETAL MACROSOMIA FOETAL MALNUTRITION FOETAL MALPOSITION FOETAL MALPRESENTATION FOETAL PLACENTAL THROMBOSIS FOETAL-MATERNAL HAEMORRHAGE GESTATIONAL DIABETES GESTATIONAL HYPERTENSION **GESTATIONAL OEDEMA** GESTATIONAL TROPHOBLASTIC DETACHMENT GLUCOSE TOLERANCE IMPAIRED IN PREGNANCY GLYCOSURIA DURING PREGNANCY HABITUAL ABORTION HAEMORRHAGE FOETAL HAEMORRHAGE IN PREGNANCY HELLP SYNDROME HETEROTOPIC PREGNANCY HIGH FOETAL HEAD HIGH RISK PREGNANCY HYDROPS FOETALIS HYPEREMESIS GRAVIDARUM HYPOTHERMIA NEONATAL **IMMINENT ABORTION** INCOORDINATE UTERINE ACTION INDETERMINATE PREGNANCY TEST RESULT INDUCED ABORTION FAILED INDUCED ABORTION HAEMORRHAGE INDUCED ABORTION INFECTION INDUCED LABOUR INJURY TO SPINAL CORD SECONDARY TO BIRTH TRAUMA INTRAPARTUM HAEMORRHAGE JAUNDICE NEONATAL LABOUR COMPLICATION LABOUR PAIN LACK OF PRENATAL CARE LACTATION NORMAL LARGE FOR DATES BABY LEUKOPENIA NEONATAL LITHOPEDION LIVE BIRTH LOCKED TWINS

CONFIDENTIAL – FOIA Exemptions Apply in U.S.

| LOW BIRTH WEIGHT BABY |
|------------------------------------------------|
| MATERNAL CANCER IN PREGNANCY |
| MATERNAL CONDITION AFFECTING FOETUS |
| MATERNAL DEATH AFFECTING FOETUS |
| MATERNAL DEATH DURING CHILDBIRTH |
| MATERNAL DISTRESS DURING LABOUR |
| MATERNAL DRUGS AFFECTING FOETUS |
| MATERNAL EXPOSURE BEFORE PREGNANCY |
| MATERNAL EXPOSURE DURING BREAST FEEDING |
| MATERNAL EXPOSURE DURING DELIVERY |
| MATERNAL EXPOSURE DURING PREGNANCY |
| MATERNAL EXPOSURE TIMING UNSPECIFIED |
| MATERNAL EXPOSURE VIA PARTNER DURING PREGNANCY |
| MECONIUM ABNORMAL |
| MECONIUM IN AMNIOTIC FLUID |
| MECONIUM INCREASED |
| MECONIUM STAIN |
| MIRROR SYNDROME |
| MISCARRIAGE OF PARTNER |
| MISSED LABOUR |
| MOLAR ABORTION |
| MORNING SICKNESS |
| MULTIGRAVIDA |
| MULTIPAROUS |
| MULTIPLE PREGNANCY |
| NEONATAL DISORDER |
| NEONATAL THYROTOXICOSIS |
| NORMAL FOETUS |
| NORMAL LABOUR |
| NORMAL NEWBORN |
| NULLI GRAVIDA |
| NULLIPAROUS |
| OBLIQUE PRESENTATION |
| OBSTRUCTED LABOUR |
| OLIGOHYDRAMNIOS |
| OMPHALORRHEXIS |
| PARITY |
| PATERNAL DRUGS AFFECTING FOETUS |
| PATERNAL EXPOSURE BEFORE PREGNANCY |
| PATERNAL EXPOSURE DURING PREGNANCY |
| PATERNAL EXPOSURE TIMING UNSPECIFIED |

| PELVIC GIRDLE PAIN |
|-------------------------------------------|
| PELVIC HAEMATOMA OBSTETRIC |
| PERINATAL BRAIN DAMAGE |
| PERINEAL REPAIR BREAKDOWN |
| PERIPARTUM CARDIOMYOPATHY |
| PERIPARTUM HAEMORRHAGE |
| PLACENTA ACCRETA |
| PLACENTA DUPLEX |
| PLACENTA PRAEVIA |
| PLACENTA PRAEVIA HAEMORRHAGE |
| PLACENTAL CALCIFICATION |
| PLACENTAL CYST |
| PLACENTAL DISORDER |
| PLACENTAL DYSPLASIA |
| PLACENTAL HYPERTROPHY |
| PLACENTAL INFARCTION |
| PLACENTAL INSUFFICIENCY |
| PLACENTAL LAKE |
| PLACENTAL NECROSIS |
| PLACENTAL POLYP |
| PLANNING TO BECOME INFERTILE |
| PLANNING TO BECOME PREGNANT |
| POLYHYDRAMNIOS |
| POLYMORPHIC ERUPTION OF PREGNANCY |
| POOR WEIGHT GAIN NEONATAL |
| POST ABORTION COMPLICATION |
| POST ABORTION HAEMORRHAGE |
| POST ABORTION INFECTION |
| POSTMATURE BABY |
| POSTNATAL GROWTH RESTRICTION |
| POSTPARTUM DISORDER |
| POSTPARTUM HAEMORRHAGE |
| POSTPARTUM STATE |
| POSTPARTUM UTERINE SUBINVOLUTION |
| PRE-ECLAMPSIA |
| PRECIPITATE LABOUR |
| PREGNANCY |
| PREGNANCY AFTER POST COITAL CONTRACEPTION |
| PREGNANCY IN HABITUAL ABORTER |
| PREGNANCY OF PARTNER |
| PREGNANCY OF UNKNOWN LOCATION |

PREGNANCY ON CONTRACEPTIVE PREGNANCY ON ORAL CONTRACEPTIVE PREGNANCY TEST PREGNANCY TEST POSITIVE PREGNANCY TEST URINE PREGNANCY TEST URINE POSITIVE PREGNANCY WITH ADVANCED MATERNAL AGE PREGNANCY WITH CONTRACEPTIVE DEVICE PREGNANCY WITH CONTRACEPTIVE PATCH PREGNANCY WITH IMPLANT CONTRACEPTIVE PREGNANCY WITH INJECTABLE CONTRACEPTIVE PREGNANCY WITH YOUNG MATERNAL AGE PREMATURE BABY PREMATURE DELIVERY PREMATURE LABOUR PREMATURE RUPTURE OF MEMBRANES PREMATURE SEPARATION OF PLACENTA PRETERM PREMATURE RUPTURE OF MEMBRANES PREVIOUS CAESAREAN SECTION **PRIMIGRAVIDA PRIMIPAROUS** PROLONGED LABOUR PROLONGED PREGNANCY PROLONGED RUPTURE OF MEMBRANES PROPHYLAXIS OF ABORTION PSEUDOMENSTRUATION NEONATAL RENAL DISORDER IN PREGNANCY RETAINED PLACENTA OR MEMBRANES RETAINED PRODUCTS OF CONCEPTION RETROPLACENTAL HAEMATOMA RISK OF FUTURE PREGNANCY MISCARRIAGE RUBELLA IN PREGNANCY RUPTURED ECTOPIC PREGNANCY SECOND TRIMESTER PREGNANCY SELECTIVE ABORTION SHORT INTERPREGNANCY INTERVAL SHOULDER DYSTOCIA SMALL FOR DATES BABY SMALL SIZE PLACENTA SOMATIC SYMPTOM DISORDER OF PREGNANCY STILLBIRTH

CONFIDENTIAL – FOIA Exemptions Apply in U.S.

SUBCHORIONIC HAEMATOMA SUBCHORIONIC HAEMORRHAGE SUPERIMPOSED PRE-ECLAMPSIA **TERM BABY** TERM BIRTH THIRD STAGE POSTPARTUM HAEMORRHAGE THIRD TRIMESTER PREGNANCY THREATENED LABOUR THYROID DYSFUNCTION IN PREGNANCY TRANSVERSE PRESENTATION TRAUMATIC DELIVERY TUBAL RUPTURE TWIN PREGNANCY UMBILICAL CORD ABNORMALITY UMBILICAL CORD AROUND NECK UMBILICAL CORD COMPRESSION UMBILICAL CORD CYST UMBILICAL CORD HAEMORRHAGE UMBILICAL CORD OCCLUSION UMBILICAL CORD PROLAPSE UMBILICAL CORD SHORT UMBILICAL CORD THROMBOSIS UMBILICAL CORD VASCULAR DISORDER UMBILICAL GRANULOMA UNINTENDED PREGNANCY UNSTABLE FOETAL LIE UNWANTED PREGNANCY **UTERINE ATONY** UTERINE CONTRACTIONS ABNORMAL UTERINE CONTRACTIONS DURING PREGNANCY UTERINE HYPERSTIMULATION UTERINE HYPERTONUS UTERINE HYPOKINESIA **UTERINE HYPOTONUS UTERINE INVERSION UTERINE IRRITABILITY** UTERINE TACHYSYSTOLE VANISHING TWIN SYNDROME VASA PRAEVIA VENOUS THROMBOSIS IN PREGNANCY WEIGHT DECREASE NEONATAL

CONFIDENTIAL – FOIA Exemptions Apply in U.S.

#### 1.11 Pulmonary venoocclusive disease associated with pulmonary oedema

The case will be included in this subgroup if it contains an event with the following MedDRA Preferred Term:

ACUTE LUNG INJURY
ACUTE PULMONARY OEDEMA
ACUTE RESPIRATORY DISTRESS SYNDROME
NEGATIVE PRESSURE PULMONARY OEDEMA
NON-CARDIOGENIC PULMONARY OEDEMA
PULMONARY CONGESTION
PULMONARY OEDEMA
PULMONARY OEDEMA
PULMONARY OEDEMA
REEXPANSION PULMONARY OEDEMA

### 1.12 Renal function impairment / acute renal failure

Cases including events denoting renal function impairment / acute renal failure are retrieved from the safety database for analysis if they contain an event PT within the MedDRA SMQ 'Acute renal failure' (narrow scope) or it contains an event with any of the following MedDRA PTs: 'Blood creatinine abnormal', 'Blood creatinine increased', 'Creatinine renal clearance abnormal', 'Creatinine renal clearance decreased', 'Glomerular filtration rate abnormal', 'Glomerular filtration rate decreased', 'Renal function test abnormal', 'Renal transplant', 'Renal tubular injury', 'Renal tubular necrosis', and 'Urine output decreased', i.e., any of the following MedDRA PTs:

| ACUTE KIDNEY INJURY |
|--------------------------------------|
| ACUTE PHOSPHATE NEPHROPATHY |
| ANURIA |
| AZOTAEMIA |
| BLOOD CREATININE ABNORMAL |
| BLOOD CREATININE INCREASED |
| CONTINUOUS HAEMODIAFILTRATION |
| CREATININE RENAL CLEARANCE ABNORMAL |
| CREATININE RENAL CLEARANCE DECREASED |
| DIALYSIS |
| FOETAL RENAL IMPAIRMENT |
| GLOMERULAR FILTRATION RATE ABNORMAL |
| GLOMERULAR FILTRATION RATE DECREASED |
| HAEMODIALYSIS |
| HAEMOFILTRATION |
| NEONATAL ANURIA |
| NEPHROPATHY TOXIC |
| OLIGURIA |
| PERITONEAL DIALYSIS |
| PRERENAL FAILURE |
| RENAL FAILURE |

CONFIDENTIAL – FOIA Exemptions Apply in U.S.

L CLIME WIND THAT DAY DAY

RENAL FAILURE NEONATAL
RENAL FUNCTION TEST ABNORMAL
RENAL IMPAIRMENT
RENAL IMPAIRMENT NEONATAL
RENAL TRANSPLANT
RENAL TUBULAR INJURY
RENAL TUBULAR NECROSIS
SUBACUTE KIDNEY INJURY
URINE OUTPUT DECREASED

# 1.13 Prostacyclin associated reactions

ARTHRALGIA
DIARRHOEA
DIZZINESS
FLUSHING
HEADACHE
MUSCULOSKELETAL PAIN
MYALGIA
NAUSEA
PAIN IN EXTREMITY
PAIN IN JAW
TEMPOROMANDIBULAR JOINT SYNDROME
VOMITING

#### 1.14 COVID-19 Infection

| ASYMPTOMATIC COVID-19 |
|-----------------------------------------------|
| CONGENITAL COVID-19 |
| CORONAVIRUS INFECTION |
| CORONAVIRUS TEST POSITIVE |
| COVID-19 |
| COVID-19 IMMUNISATION |
| COVID-19 PNEUMONIA |
| COVID-19 PROPHYLAXIS |
| COVID-19 TREATMENT |
| EXPOSURE TO SARS-COV-2 |
| MULTISYSTEM INFLAMMATORY SYNDROME IN CHILDREN |
| OCCUPATIONAL EXPOSURE TO SARS-COV-2 |
| POST-ACUTE COVID-19 SYNDROME |
| SARS-COV-2 ANTIBODY TEST POSITIVE |
| SARS-COV-2 CARRIER |
| SARS-COV-2 RNA DECREASED |
| SARS-COV-2 RNA FLUCTUATION |

CONFIDENTIAL – FOIA Exemptions Apply in U.S.

| SARS-COV-2 RNA INCREASED |
|--------------------------------------|
| SARS-COV-2 SEPSIS |
| SARS-COV-2 TEST FALSE NEGATIVE |
| SARS-COV-2 TEST POSITIVE |
| SARS-COV-2 VIRAEMIA |
| SUSPECTED COVID-19 |
| VACCINE DERIVED SARS-COV-2 INFECTION |

Status: Approved, Date: 2 May 2022